

#### STATISTICAL REPORTING AND ANALYSIS PLAN

Impact of a Nutritional supplement on Bone turnover markers in Indian healthy premenopausal women (25-45 yrs; inclusive) after 6 months of intervention: A randomised double blind controlled trial

**Protocol Number:** 207192

Phase: N/A

Property of GSK Consumer Healthcare
Confidential
May not be used, divulged, published or otherwise disclosed
without the consent of GSK
Template Version Effective: 15-Jul-2017


## **Document History**

| Document | Version Date | Summary of Changes (New analysis or Change in planned analysis) |
|---|---|---|
| Original Analysis Plan | 13-February-2018 | Not applicable (N/A) |
| Final Statistical Reporting and Analysis Plan Amendment Version 1.0 | 13-April-2018 | <ol> <li>Section 1.4 is updated for the typo.</li> <li>Seven day dietary intake assessment information is collected at baseline and at Month 6 (visit 6) as per Protocol and eCRF. However, this information was missed while developing the RAP. Therefore, Section 4.6 has been updated to include this information as well as one summary table and one listing.</li> <li>Section 4.4.1.2 is updated with 97.5 % CI. This is because 95% CI was as per protocol just to correct the same RAP section is updated along with tables 14.2.2.2, 14.2.3.2 and 14.2.2.2a, 14.2.3.2a.</li> <li>Section 5, updated to document the changes from the protocol and RAP.</li> <li>The analysis population on template for Table 14.2.2.2a was planned as safety however, there was a typo and it is now updated from ITT to Safety population.</li> <li>The title and the format of the laboratory shift tables (Table 14.3.5.3 till 14.3.12) updated since it will be helpful for the programmers and reviewers</li> <li>Section 4.7.2 is updated since vendor laboratory confirmed that for the following tests, normal ranges will not be available: Serum Cross-Linked C-Telopeptide of Type 1 Collagen, Ratio of Carboxylated to Under-Carboxylated Osteocalcin, Urinary C-Telopeptide of Type 1 Collagen, Serum Vitamin D (using 25-OH D3), Urinary Calcium/Creatinine Ratio and Serum Folate. The shift tables related to these parameters are deleted and programming note is added for the listings.</li> </ol> |
| | | <ul> <li>8. Added Table 14.2.20.1, for the summary of dietary assessment</li> <li>9. Deleted two rows from the Table 14.3.1.3 "Treatment Emergent Adverse Events by System</li> </ul> |
| | | Organ Class, Preferred Term and Severity since those are not required in this table. |
| | | 10. From listing 16.2.9.3 three columns (Blood collection date and time, kit number and cold chain start time,) have been deleted since these are |

| Document | Version Date | Summary of Changes (New analysis or Change in planned analysis) |
|---|---|---|
| | | same for all blood related parameters and not specific for the HB assessment. Also a footnote is added to explain the meaning of assessment performed (yes/no). 11. Updated the title of all the tables related to the statistical analysis to reflect that the analysis is performed on the change from baseline response variable. 12. Fourth column name in the Listing 16.2.5.1 updated to adjust the space and programming note added. |
| Final Statistical Reporting and Analysis Plan Addendum Version 1.0 | 01-June-2018 | <ol> <li>Added Section 4.3.1.1 which details a study product compliance summary by categories 0-3 months and 3-6 months. This is added to check if the difference in compliance could be linked to the difference in the primary parameter results between Month 3 and Month 6.</li> <li>Added statistical model for the sensitivity analysis for log-transformed s-CTX1 in Section 4.4.1.2</li> <li>Added Section 4.4.1.4 which details a subgroup ANCOVA analysis on s-CTX1 change from baseline by age strata at Month 3 and Month 6. This analysis is added to check if age has an impact on the treatment effect.</li> <li>Added statistical model for the sensitivity analysis for log-transformed data for the secondary endpoints in Section 4.4.2.</li> <li>Added Section 4.6.1 which details an ANCOVA analysis on the change from baseline of each dietary intake parameter assessment. This is added to assess if significant changes in dietary intake can be linked to change in primary endpoints at Month 6.</li> <li>Details added to Section 5 summarizing the above ad-hoc analyses with justification and timing.</li> </ol> |
| Final Statistical<br>Reporting and Analysis<br>Plan Addendum<br>Version 2.0 | 23-July-2018 | Added section 4.6.2 which details further post hoc analysis for a new lab parameter urine CTX-1 over creatinine ratio (CTX1CR). This variable was not previously specified in the protocol or previous versions of the analysis plan. |

Amendments incorporate all revisions to date.

| Ta | | f conteinment His | <b>nts</b><br>tory | 2 |
|---|---|---|---|---|
| | | | nts | |
| 1 | | | Ley Protocol Information | |
| | 1.1 | • | Design | |
| | 1.2 | • | Objectives | |
| | 1.3 | • | ents | |
| | 1.4 | Sample | e Size Calculation | 9 |
| 2 | Planı | _ | /ses | |
| | 2.1 | Interim | Analysis | 11 |
| | 2.2 | | analyses | |
| 3 | Cons | onsiderations for data analyses and Data Handling Conventions | | |
| | 3.1 | | ne Definition | |
| | 3.2 | Subgro | pups/Stratifications | 12 |
| | 3.3 | Centers | s Pools | 12 |
| | 3.4 | Time p | oints and Visit Windows | 12 |
| 4 | Data | Data Analysis | | |
| | 4.1 | Popula | tions for Analysis | 12 |
| | | 4.1.1 | Subject Disposition | 12 |
| | | 4.1.2 | Protocol Deviations | 13 |
| | | 4.1.3 | Analysis Populations | 14 |
| | 4.2 | Subject | t Demographics and Other Baseline Characteristics | 15 |
| | | 4.2.1 | Demographic Characteristics | 15 |
| | | 4.2.2 | General Medical History | 15 |
| | | 4.2.3 | Characteristics of Disease | 15 |
| | 4.3 | 4.3 Treatments (Study Product, Rescue Medication, other Concomitant Therapies, Compliance) | | 15 |
| | | 4.3.1 | Study Product Compliance and Exposure | 15 |
| | | 4.3.2 | Prior and Concomitant Medication | 17 |
| | 4.4 | Analys | is of Efficacy | 17 |
| | | 4.4.1 | Primary Efficacy Endpoint | |
| | | 4.4.2 | Secondary Efficacy Variables | 20 |
| | | 4.4.3 | Handling of Missing Values/Censoring/Discontinuations | 21 |

| | 4.5 | Analys | is of Secondary Objectives | 22 |
|-----|------|------------|----------------------------------------------|----|
| | | 4.5.1 | Efficacy (Secondary) | 22 |
| | 4.6 | Explora | atory Analysis | |
| | | 4.6.1 | Dietary Intake Assessment Post hoc Analyses | |
| | | 4.6.2 | Further Post hoc Analysis | 23 |
| | 4.7 | Analys | is of Safety | |
| | | 4.7.1 | Adverse Events and Serious Adverse Events | 24 |
| | | 4.7.2 | Laboratory Tests | 24 |
| | | 4.7.3 | Vital Signs | 25 |
| | | 4.7.4 | Findings on Physical Examination | |
| | | 4.7.5 | Other Safety Variables | 25 |
| | 4.8 | Analys | is of Other Variables | |
| | | 4.8.1 | Quality of Life | |
| | | 4.8.2 | Patch Adhesion Performance | 26 |
| 5 | Chan | ges to the | e Protocol Defined Statistical Analysis Plan | 26 |
| Att | | _ | of Data Displays | |
| 6 | | | Tables, Figures and Listings | |

## **Abbreviation**

| Abbreviation | Term |
|---|---|
| AE | Adverse Event |
| ALP | Alkaline Phosphatase |
| BDRM | Blinded Data Review Meeting |
| BSAP | Bone Specific Alkaline Phosphatase |
| Ca | Calcium |
| CI | Confidence Interval |
| c-OC | Carboxylated osteocalcin |
| c-OC/uc-OC | Ratio of carboxylated osteocalcin to under carboxylated osteocalcin |
| GSK CH | GlaxoSmithKline Consumer Healthcare |
| ITT | Intent-To-Treat |
| MedDRA | Medical Dictionary for Regulatory Activities |
| P | Phosphorous |
| PP | Per-Protocol |
| PT | Preferred Term |
| s-CTX-1 | Serum C-terminal cross-linking telopeptide of type I collagen |
| s-NTX-1 | Serum N-terminal cross-linking telopeptide of type I collagen |
| s-P1NP | Serum N-terminal propeptide of type I procollagen |
| SD | Standard Deviation |
| SE | Standard Error |
| Se | Selenium |
| SI | International System of units |
| SOC | System Organ Class |
| TEAE | Treatment Emergent Adverse Event |
| 25 OH D3 | 25 Hydroxycalciferol |
| uc-OC | Under carboxylated osteocalcin |
| u - CTX-1 | Urinary C-terminal telopeptide of type I collagen |
| Zn | Zinc |

The purpose of this Statistical Reporting and Analysis Plan is to describe the planned analyses and outputs to be included in the Clinical Study Report for Protocol 207192.

## 1 Summary of Key Protocol Information

Change in life style, dietary habits and environment is known to have significant effect on women's physiology and bones are not spared from the impact. In post-menopausal women, the prevalence of low bone mineral density (BMD), its association to fracture risk and efficacy of pharmacologic therapy to reduce the risk of fractures are well established. The World health Organization (WHO) criteria for diagnosing Osteopenia and Osteoporosis are also based on epidemiological data obtained in post-menopausal women and the treatment guidelines are also targeted for post-menopausal women.

GSK India consumer healthcare has developed a customized nutritional supplement product designed to improve bone health in Indian women. The purpose of this study is to assess efficacy of the supplement on bone health. Two reference bone turnover markers serum C-telopeptide of type I collagen (s-CTX-1) and N-terminal propeptide of type I procollagen (PINP) recommended by International Osteoporosis foundation will be utilized to assess the impact of Women's Horlicks in Indian health pre-menopausal women aged group 25-45 years (inclusive), following six months supplementation.

## 1.1 Study Design

This is a double blind, single-centre, two-arm, parallel group, randomized-controlled, in 25-45 year old menopausal women. This subject will be stratified by age bands with an aim to recruit a target ratio of 50% in the  $\geq$ 25- $\leq$ 35 years age band and 50% in the  $\geq$ 35- $\leq$ 45 years age band with a minimum of 40% of either age band.

The trial will have two groups.

Test product (Group 1): Protein rich beverage powder fortified with MMN

Reference product (Group 2): Low protein non-fortified iso-caloric beverage powder

## 1.2 Study Objectives

| Objectives | Endpoints |
|---|---|
| Primary Objective | Primary Endpoint |
| <ul> <li>To compare the changes in Bone Resorption<br/>marker: serum C-telopeptide of type 1<br/>collagen (s-CTX-1) at end line 6 months<br/>from baseline in test and control groups</li> </ul> | Change from baseline in s-CTX-1 at 6 months |
| <ul> <li>To compare the changes in the ratio of<br/>carboxylated (c-OC) to under-carboxylated</li> </ul> | Change from baseline in the ratio of c-OC to uc-OC at 6 months |

| Objectives | Endpoints |
|---|---|
| Osteocalcin (uc-OC) at end line 6 months | |
| from baseline in test and control groups | |
| Secondary Objectives | Secondary Endpoints |
| Efficacy | |
| <ul> <li>To compare the changes in Bone Resorption<br/>marker: serum C-telopeptide of type 1<br/>collagen (s-CTX-1) at mid line 3 months<br/>from baseline in test and control groups</li> </ul> | Change from baseline in s-CTX-1 at 3 months |
| <ul> <li>To compare the changes in the ratio of<br/>carboxylated (c-OC) to under-carboxylated<br/>Osteocalcin (uc-OC) at mid line 3 months<br/>from baseline in test and control groups</li> </ul> | Change from baseline in the ratio of c-OC to uc-OC at 3 months |
| <ul> <li>To compare the changes in Bone Resorption<br/>marker: urinary CTX -1 at mid line 3 months<br/>and end line 6 months from baseline in test<br/>and control groups</li> </ul> | Change from baseline in urinary CTX-1 at 3 months and at 6 months |
| <ul> <li>To compare the changes in Bone Resorption<br/>marker: serum N-terminal telopeptide of type<br/>1 collagen (s-NTX-1) at mid line 3 months<br/>and at end line 6 months from baseline in<br/>test and control groups</li> </ul> | Change from baseline in s-NTX-1 at 3 months and at 6 months |
| <ul> <li>To compare in bone formation marker serum<br/>procollagen type 1 N-terminal propeptide (s-<br/>P1NP), bone specific alkaline phosphatase<br/>(BSAP) at baseline, at mid line 3 months<br/>and at end line 6 months in test and control<br/>groups</li> </ul> | Change from baseline in s-P1NP and BSAP at 3 months and at 6 months |
| <ul> <li>To compare calcium status using s-PTH and<br/>urinary calcium, serum Ca, P and total<br/>alkaline phosphatase (ALP) at mid line 3<br/>months and end line 6 months to see<br/>change in level from baseline in both the<br/>groups</li> </ul> | Change from baseline in s-PTH and urinary calcium, serum Ca, P and total alkaline phosphatase (ALP) at 3 months and at 6 months |
| To compare the changes in Vitamin D status using serum 25-hydroxycholecalciferol (25 OH D3) at mid line 3 months and end line 6 months from baseline in test and control groups | Change from baseline in 25-hydroxycholecalciferol (25 OH D3) at 3 months and 6 months |
| To compare the changes in micronutrient profile status sing serum Se, Folic acid, B12 and plasma Zn and B6 at mid line 3 months and end line 6 months from baseline in test and control groups | Change from baseline in Se, Folic acid, B12 and plasma Zn and B6 status at 3 months and 6 months |
| Exploratory Objectives | Exploratory Endpoints |

| Objectives | Endpoints |
|---|---|
| To compare the changes in growth markers<br>IGF-1 at mid line 3 months and end line 6<br>months from baseline in test and control<br>groups | Change from baseline in IGF-1 at 3 months and 6 months |

#### 1.3 Treatments

The study products are as follows:

| | Test Product 1 | Reference Product 1 |
|---|---|---|
| Product Name | Cereal based fortified<br>Beverage (Proprietary food) | Low protein non fortified isocaloric beverage |
| Product Formulation<br>Code (MFC) | CCI | CCI |
| Dose | 60 grams daily in two divided doses | 60 grams daily in two divided doses |
| Route of Administration | Oral | Oral |
| Dosing Instructions | 30 grams powder made up in 200 mL water, administered twice daily | 30 grams powder made up in 200 mL water, administered twice daily |

### 1.4 Sample Size Calculation

The first primary objective for this study is changes in s-CTX-1 levels. Naylor et al. (2015) used bone turnover markers to identify women who responded to bisphosphonate treatment for osteoporosis. The change in CTX with risedronate (above the effect of the calcium and vitamin D supplement) was 30%. Thus, we can say that a 30% reduction has been shown to be associated with a reduction in fractures. Hence, a reduction of 20% in test product as compared to placebo could be considered as a clinically significant difference.

Estimates of mean s-CTX-1 and variability from Kruger et al, 2006 were as follows:

Estimates of s-CTX-1 and variability from Kruger et al, 2006 (Mean  $\pm$  Standard Deviation [SD]1)

| Endpoint | | Test Product | Control Product |
|----------|-------------------------|-------------------|------------------|
| | Baseline | $0.45 \pm 0.166$ | $0.44 \pm 0.032$ |
| CTX-1 | Post-Baseline (Week 16) | $0.30 \pm 0.094$ | $0.46 \pm 0.092$ |
| | Change from baseline | $-0.15 \pm 0.144$ | $0.02 \pm 0.142$ |

1: Standard Error (SE) values were reported in the paper. SD was calculated as SE\*SQRT (N).

SD values for change from baseline were not reported in the paper. These were calculated using following formula considering correlation coefficient between baseline and post-baseline values as 0.5:

$$SD_{E,change} = \sqrt{SD_{E,base line}^2 + SD_{E,final}^2 - (2 \times Corr \times SD_{E,base line} \times SD_{E,final})}$$

SDE, change = SD for change from baseline

SDE,baseline = SD for baseline

SDE, final = SD for post-baseline

Corr = correlation coefficient between baseline and final values

Considering similar baseline values and 20% clinically relevant decrease in test product (lower values are better) from baseline, -0.09 will be used as change from baseline value in test product. This gives a treatment difference of -0.11.

Based on the above estimates of treatment difference and taking the larger estimate for variability (SD = 0.144), to be able to achieve 90% power, 44 participants per treatment arm (Total = 88) will be required to complete the study. This assumes 2.5% level of significance (two tailed t-test).

To allow for 20% drop-out rate, a total of 54 participants (Total = 108) will be randomized per treatment arm.

The co-primary objective for this study is changes in (c-OC/uc-OC) levels. From Binkley et al. the following data related to the end point was received.

From the estimates of %uc-OC, and Total OC from Binkley et al (Mean), the estimates of c-OC have been calculated. From the available data the following table has been tabulated.

| Endpoint | | Test Product | Control Product |
|------------|------------------------|--------------|-----------------|
| | Baseline | 11.7206 | 11.96 |
| c-OC/uc-OC | Post-Baseline (Week 2) | 31.806 | 18.60 |
| | Change from baseline | 20.14 | 7.53 |

Considering the delta value as 12.5 and the SD as 13 using Taylor series expansion the sample size to be able to achieve 90% power, 30 participants per treatment arm (Total = 60) will be required to complete the study. This assumes 2.5%% level of significance (two tailed t-test).

To allow for 20% drop-out rate, a total of 36 participants (Total = 72) will be randomized per treatment arm.

However, the sample size for the first primary end point is larger so the sample size will be required for this study is 108 in total.

The sample size is based on the primary endpoint. No sample size considerations have been taken into account for secondary objectives.

Approximately 135 participants will be screened to randomize approximately 108 participants in order to obtain 88 participants completing the study.

Following assumptions have been taken for sample size estimation:

Estimates of s-CTX-1 will be similar in Indian Women as compared to New Zealand Population (Kruger et al, 2006). Product used in Kruger et al, 2006 and in the proposed study will provide similar estimates of s-CTX-1.

Values at 6 months in the proposed study will be similar to values at 4 months from Kruger et al. 2006.

Women 25-35 years old will have similar estimates of s-CTX-1 as 36-45 years old from Kruger et al

Vitamin K supplementation reduces serum concentrations of under carboxylated osteocalcin in healthy young and elderly adults from Binkley et al.

## 2 Planned Analyses

### 2.1 Interim Analysis

No interim analysis is planned.

## 2.2 Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and database has been locked.
- 3. All criteria for un-blinding the randomisation codes have been met and the randomisation codes have been distributed.

## 3 Considerations for data analyses and Data Handling Conventions

#### 3.1 Baseline Definition

For all endpoints the baseline value will be the latest pre-dose assessment with a non-missing value. Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.

### 3.2 Subgroups/Stratifications

In this study subjects will be stratified by their age groups defined as follows:

- Stratum 1: Age  $\geq$  25 years; age < 35 years
- Stratum 2: Age  $\geq$  35 years; age  $\leq$  45 years

For details on subgroup analyses please refer to section 4.1.4.

#### 3.3 Centers Pools

Since this is a single center study, pooling of centers is not applicable.

#### 3.4 Time points and Visit Windows

The time points and visits for this study are defined in the section "Schedule of Events" of the protocol. Any deviation from the study schedule will be reviewed case-by-case basis to determine whether the data should be excluded from the Per-Protocol (PP) population. A time window non-compliance listing will be produced for the Blinded Data Review Meeting (BDRM) only.

## 4 Data Analysis

Data analysis will be performed by InVentiv Health. The statistical analysis software used will be SAS Studio version 9.4 or higher.

Prior to database closure a BDRM will be conducted in which various aspects of the trial will be discussed and agreed.

Unless otherwise described below, all listings will be produced for All Randomized Subjects.

#### 4.1 Populations for Analysis

#### 4.1.1 Subject Disposition

Screen failures are defined as subjects who consent to participate in the clinical study but are not subsequently randomized. A summary of the number of subjects screened and the number of screen failures with reasons why subjects were not randomized will be presented (Table 14.1.1). For the summary of screen failure subjects the percentages will be based on total number of screened subjects.

GlaxoSmithKline Consumer Healthcare 

Subject disposition will also be summarized by treatment group and overall as the number and percentage of subjects who complete the study, with the number who discontinue broken down by reason for discontinuation (Table 14.1.1). The table will also summarize the number and percent of subjects assigned to each analysis population (refer to Section 4.1.3). The percentage will be based on total number of subjects randomized in each product and overall.

Subject disposition including the subject status (completer, Yes/No), demographic data (age and race), screening date, study product start date and time, the duration in the study or trial [(date/time of completion/withdrawal minus date of first dose administration)+1] and the specific reason for discontinuation, will be listed for randomized subjects (Listing 16.2.1.1.1) by product group.

Subject disposition information for non-randomized subjects will include subject number, demographic information (age and race), screening date, reason for screen failure and details if any regarding the reason for screen failure (Listing 16.2.1.1.2).

#### 4.1.2 Protocol Deviations

Protocol deviations will be tracked by the study team throughout the conduct of the study. Data will be reviewed prior to un-blinding and closure of the database to ensure all important deviations are captured and categorized. Subjects with major protocol deviations (defined below) will be excluded from the PP population.

Major deviations of the protocol procedures identified as liable to influence the efficacy outcomes of the study may include, but will not be necessarily limited to the following:

- Violation of inclusion or exclusion criteria
- Significant non-compliance with assigned treatment
- Efficacy assessments outside the specified time windows
- Use of prohibited treatment or medication before or during the study
- Any other reason identified which may affect the efficacy assessments

The number and percentage of subjects with any major protocol deviations will be presented by product group and overall (Table 14.1.2) and listed in Listing 16.2.2.1. Any minor protocol deviations will be listed similarly (Listing 16.2.2.2).

#### 4.1.3 Analysis Populations

In this study the following analysis populations are defined:

| Population | Definition / Criteria | <b>Analyses Evaluated</b> |
|---|---|---|
| Randomized Population | All subjects who are randomized and<br>may or may not have received the<br>study product | Disposition |
| Safety Population | <ul> <li>All subjects who are randomized and have received at least one dose of study product.</li> <li>The safety population will be analysed as per product received.</li> </ul> | Safety |
| Intent-to-treat (ITT) Population | All subjects in the safety population who have at least one post product co-primary efficacy assessment (either s-CTX-1 or ratio of carboxylated (c-OC) to under-carboxylated Osteocalcin (uc-OC). | Efficacy |
| PP Population | A subset of the ITT population excluding subjects with major protocol deviations. Depending on the nature of the major protocol deviation and impact on the efficacy variable(s), subjects will be either wholly excluded from the PP population or only partially excluded from the PP analyses. This will be determined on a case-by-case basis. | Efficacy |

**NOTES :** Please refer to Attachment 1: List of Data Displays which details the population to be used for each displays being generated.

Subjects excluded from any of the analysis populations will be listed in Listing 16.2.3.1, with the reason for exclusion.

The primary population for assessment of efficacy will be the ITT population. A PP analysis will be performed for the co-primary endpoints only if 10% or more ITT subjects are excluded from the PP population.

### 4.2 Subject Demographics and Other Baseline Characteristics

#### 4.2.1 Demographic Characteristics

Descriptive statistics (number of subjects [n], mean, median, standard deviation [SD], minimum and maximum) for the continuous variables and frequency (n) and percentages (%) for categorical variables will be provided for demographic variables. The demographic and baseline data will include age (years), sex, race, weight (kg), height (cm) and body mass index (kg/m²). The number and percentage of subjects in each stratum will also be presented.

All demographic information will be tabulated by product group and overall in Table 14.1.4.1 for the Safety population, Table 14.1.4.2 for the ITT population, Table 14.1.4.3 for the PP population and listed in Listing 16.2.4.1.

#### 4.2.2 General Medical History

Medical history and current medical conditions will be listed in Listing 16.2.4.2, with start date and end date or ongoing.

#### 4.2.3 Characteristics of Disease

Not Applicable.

# 4.3 Treatments (Study Product, Rescue Medication, other Concomitant Therapies, Compliance)

#### 4.3.1 Study Product Compliance and Exposure

The descriptive summary of total number of dispensed, consumed and returned sachets will be presented by product group and overall for all subjects in ITT population (Table 14.2.1.1). The data used for these summaries will be taken directly from the eCRF recorded data. These are the following things which will be re-calculated due to some data discrepancies observed in data capturing –

Percentage compliance with study product will be computed for each subject at each visit as: (Actual number of sachets consumed / expected number of sachets consumed) X 100 where:

GlaxoSmithKline Consumer Healthcare 

actual total number of sachets consumed = (number of sachets dispensed –number of sachets unconsumed returned)

expected number of sachets consumed = (2 sachets X number days between visits).

For the by visit compliance calculation the number of days between visits will be between two consecutive visits. For the overall compliance calculation the number of days between visits will be between visit 2 and visit 6.

Percentage overall study product compliance across the entire study duration will be computed as:

(Total number of actual sachets consumed/total number of expected sachets consumed) X 100.

The "actual number of sachets consumed" will not use the number of returned empty sachets reported on the eCRF, as some sachets may be consumed but not returned by subjects.

Summary statistics of overall study product compliance will be presented by product group (Table 14.2.1.1). Subject will be considered non-compliant if the compliance calculation is less than 80% of the total amount of recommended dose. The number of compliant and non-compliant subjects will be summarized by frequency count and percentage (Table 14.2.1.1). The date/time of product administration, exposure and study product compliance will also be listed in Listing 16.2.5.1.

Exposure to the study product in days will be calculated as date of last study product administration minus date of first study product administration +1. Exposure to the study product will be summarized descriptively by product group and overall for all subjects in ITT population in the same table mentioned above and will be listed in Listing 16.2.5.1.

Study product compliance will be reviewed during then BDRM and a listing will be produced for evaluation of protocol deviations. Study product non-compliance regarded to influence the primary efficacy endpoints will be excluded from PP analysis. Any subject and/or time point excluded from PP analysis will be clearly documented in population definition document.

#### 4.3.1.1 Study Product Compliance Post hoc Analyses

Summary statistics of the overall study product compliance between 0-3 months and 3-6 months will be presented by product group (Table 14.2.1.1a). The categories will be defined in the following ways –

Category 1: 0 - 3 months: This category will assess the compliance between Visit 2 to Visit 4, where the compliance assessment will be calculated using Visit 3 and Visit 4.

GlaxoSmithKline Consumer Healthcare Confidential


Category 2: 3 - 6 months: This category will assess the compliance between Visit 4to Visit 6 where the compliance assessment will be calculated using Visit 5 and Visit 6.

For the overall compliance calculation the number of days between visits will be between visit 2 and visit 4 for category 1 and between visit 4 and visit 6 for category 2 respectively.

#### 4.3.2 Prior and Concomitant Medication

Prior or concomitant medication and concomitant non-drug treatment/procedure taken by or administered to a subject will be recorded in the case report form. The prior and concomitant medications will be coded using an internal validated medication dictionary, GSK Drug.

Prior medications are defined as the medications which started and stopped before first administration of study product. If the stop date is unknown or incomplete and medication cannot be considered as stopped prior to first administration of study product then the medication will be considered as a concomitant medication.

Concomitant medications are defined as medications which started before the first administration of study product and continued during the study or medication taken between the date of first dose and last dose of study product.

Unknown dates will not be imputed, however if the start date is unknown, then it will be assumed to concomitant medication, unless the partial start date or stop date indicates differently.

Prior and concomitant medications/non-drug therapies will be listed by subject, with drug name, GSK drug synonym, indication, route, dose, frequency, start date, end date or ongoing and start day of medication (relative to first dose of study product) (Listing 16.2.5.2 and Listing 16.2.5.3).

#### 4.4 Analysis of Efficacy

#### 4.4.1 Primary Efficacy Endpoint

#### 4.4.1.1 Primary Efficacy Endpoint Definition

The primary efficacy variables of the study are:

- Change from baseline in bone resorption marker s-CTX-1 after 6 months.
- Change from baseline in the ratio of c-OC to uc-OC (c-OC/uc-OC) after 6 months.

GlaxoSmithKline Consumer Healthcare Confidential


#### 4.4.1.2 Statistical Hypothesis, Model, and Method of Analysis

The primary success criteria is to observe a statistically significantly greater reduction in s-CTX-1 for the test product than the reference product or to observe a statistically significantly greater increase in c-OC/uc-OC for the test product than the reference product, after 6 months of treatment

The hypotheses for the co-primary endpoints are:

#### • s-CTX-1:

H<sub>0P</sub>: There is no difference in mean change from baseline in bone resorption marker s-CTX-1 between reference product and test product after 6 months of treatment

H<sub>0P1</sub>: There is a difference in mean change of baseline in bone Resorption marker s-CTX-1 between reference product and test product after 6 months of treatment

#### • c-OC/uc-OC:

H<sub>0CP</sub>: There is no difference in mean change from baseline in the c-OC/uc-OC between reference product and test product after 6 months of treatment

H<sub>0CP1</sub>: There is a difference in mean change from baseline in the c-OC/uc-OC between reference product and test product after 6 months of treatment

Summary statistics (n, mean, SD, SE, median, minimum and maximum) by product group and visit of the observed and change from baseline values will be provided for both s-CTX-1 and c-OC/uc-OC (Table 14.2.2.1 and 14.2.3.1, Listing 16.2.6.1 and 16.2.6.2).

The co-primary efficacy variables will be analysed using the analysis of covariance (ANCOVA). The ANCOVA will have product group, age strata as fixed effects and the corresponding baseline value (baseline value of s-CTX-1 and/or c-OC/uc-OC as appropriate) as covariate. Adjusted means, 95% confidence intervals (CIs), within product p-values for each product group, product group difference, SE, 97.5% confidence interval of the difference and the between-product p-values based on the statistical model described above will also be presented (Table 14.2.2.2, 14.2.3.2). Statistical tests to compare treatments will be two-sided and will employ a level of significance of  $\alpha = 0.025$ .

The setting of the significance level of 0.025 for these 2 co-primary endpoints will ensure that the overall significance level for the primary endpoint is less than or equal to 0.05.

Assumptions of normality and homogeneity of variances in the ANCOVA model will be evaluated after study un-blinding. If violations are observed then the following will be performed as a post-hoc sensitivity analysis and results will be compared with primary analysis results:

1. Suitable data transformations will be tried to achieve the assumptions.

2. If suitable transformations cannot be found, then the non-parametric Van Elteren tests will be performed adjusting for age strata for each endpoint.

To visually inspect the treatment effect of s-CTX-1 and c-OC/uc-OC, plots across time (Baseline, Month 3 and Month 6) will be displayed with LSmeans and  $\pm$  SE bars which will be obtained from the ANCOVA analysis. The plot will display a different symbol line for each treatment group (Figure 14.2.2.1 and 14.2.3.1).

As post-hoc sensitivity analysis s-CTX-1 will be log-transformed (natural logarithm) and the log-transformed data will be analysed using ANCOVA model with product group, age strata as fixed effects and the corresponding log-transformed baseline value as a covariate. The interpretation of the data will be based on the geometric mean ratio and 95% confidence interval and p-value (Table 14.2.2.2c).

#### 4.4.1.3 Supportive Analyses

A supportive analysis will be performed on the co-primary variables of s-CTX-1 and c-OC/uc-OC using the statistical methodology described in Section 4.4.1.2 on all subjects in PP population, if more than 10% of the subjects in the ITT population are excluded from the PP population (Table 14.2.2.3, 14.2.3.3).

A sensitivity analysis using multiple imputations to handle missing data will be performed for each of the primary efficacy endpoints on the safety population (see Section 4.4.3).

#### 4.4.1.4 Post hoc Analyses

Summary statistics (n, mean, SD, SE, median, minimum and maximum) by product group, age strata and visit of the observed and change from baseline values will be provided for s-CTX-1 (Table 14.2.2.1a).

A post hoc subgroup ANCOVA analysis will be performed on one of the co-primary variables s-CTX-1 by age strata (as defined in section 3.2) using ITT population. The ANCOVA model will have product group, strata and (product \* strata) interaction as fixed effects and the corresponding baseline value (baseline value of s-CTX-1) as covariate. Adjusted means, 95% confidence intervals (CIs), within product p-values for each product group, product group difference, SE, 95% confidence interval of the difference and the between-product p-values based on the statistical model described above will also be presented (Table 14.2.2.2b). Statistical tests to compare treatments will be two-sided and will employ a level of significance of  $\alpha = 0.05$ .

#### 4.4.2 Secondary Efficacy Variables

The secondary efficacy variables are:

- Change from baseline in Serum C-telopeptide of type I collagen (s-CTX-1) after 3 months of treatment
- Change from baseline in Ratio of Carboxylated Osteocalcin to Under Carboxylated Osteocalcin (c-OC/uc-OC) after 3 months of treatment
- Change from baseline in Urinary C-telopeptide of type I collagen (u- CTX-1) after 3 and 6 months of treatment
- Change from baseline in Serum N-terminal telopeptide of type –I collagen (s-NTX-1) after 3 and 6 months of treatment
- Change from baseline in Serum procollagen type I N-terminal propeptide (s-P1NP) after 3 and 6 months of treatment
- Change from baseline in Bone Specific Alkaline Phosphatase (BSAP) after 3 and 6 months of treatment
- Change from baseline in Serum Parathyroid Hormone (s-PTH) after 3 and 6 months of treatment
- Change from baseline in Urinary Calcium/Creatinine ratio (USING CREATININE IN SPOT TEST TO NORMALISE) after 3 and 6 months of treatment
- Change from baseline in Serum Calcium (Ca) after 3 and 6 months of treatment
- Change from baseline in Serum Phosphorus (P) after 3 and 6 months of treatment
- Change from baseline in Serum Alkaline phosphatase (ALP)after 3 and 6 months of treatment
- Change from baseline in 25 Hydroxycalciferol (25 OH D3) after 3 and 6 months of treatment
- Change from baseline in Serum Selenium (Se) after 3 and 6 months of treatment
- Change from baseline in Plasma Zinc (Zn) after 3 and 6 months of treatment
- Change from baseline in Serum Folic acid after 3 and 6 months of treatment
- Change from baseline in Plasma B6 after 3 and 6 months of treatment
- Change from baseline in Serum B12 after 3 and 6 months of treatment

Summary statistics (n, mean, SD, SE, median, minimum and maximum) by product group and visit of the observed and change from baseline values will be provided for all secondary efficacy variables in Section 4.2.2.

GlaxoSmithKline Consumer Healthcare Confidential
Page **20** of **73** 

Each of these secondary efficacy variables will be analyzed using the ANCOVA. The ANCOVA will have product group, age strata as fixed effects and the corresponding baseline value as covariate. Adjusted means, 95% confidence intervals, within product p-values for each product group, product group difference, SE, 95% confidence interval of the difference and the between-product p-values based on the statistical model described above will also be presented (Table 14.2.4.2, Table 14.2.5.2, 14.2.6.2,14.2.7.2,14.2.8.2, 14.2.9.2, 14.2.10.2, 14.2.11.2,14.2.12.2, 14.2.13.2, 14,2.14.2,14.2.15.2, 14.2.16.2, 14.2.17.2, 14.2.18.2). Statistical tests to compare treatments will be two-sided and will employ a level of significance of  $\alpha = 0.05$ .

Assumptions of normality and homogeneity of variances in the ANCOVA model will be evaluated after study un-blinding. If violations are observed then the following will be performed as a post-hoc sensitivity analysis and results will be compared with primary analysis results:

- 1. Suitable data transformations will be tried to achieve the assumptions.
- 2. If suitable transformations cannot be found, then the non-parametric Van Elteren tests will be performed adjusting for age strata for each endpoint.

To visually inspect the treatment effect of s-CTX-1 and c-OC/uc-OC, plots across time (Baseline, Month 3 and Month 6) will be displayed with LSmeans and ± SE bars which will be obtained from the ANCOVA analysis. The plot will display a different symbol line for each treatment group (Figure 14.2.4.1, 14.2.5.1, 14.2.6.1, 14.2.7.1, 14.2.8.1, 14.2.9.1, 14.2.10.1, 14.2.11.1, 14.2.12.1, 14.2.13.1, 14.2.14.1, 14.2.15.1, 14.2.16.1, 14.2.17.1, 14.2.18.1).

As post-hoc sensitivity analysis Urinary Calcium/Creatinine ratio will be log-transformed (natural logarithm) and the log-transformed data will be analysed using ANCOVA model with product group, age strata as fixed effects and the corresponding log-transformed baseline value as a covariate. The interpretation of the data will be based on the geometric mean ratio and 95% confidence interval and p-value (Table 14.2.9.2a).

#### 4.4.3 Handling of Missing Values/Censoring/Discontinuations

Missing data will not be replaced or imputed. Subjects who withdraw from the study prematurely will be included in the statistical analyses up to the point of discontinuation.

As a part of sensitivity analysis a multiple imputation technique for imputing missing data will be conducted on ANCOVA analysis for each of the primary efficacy endpoints on the safety population. This will help to assess the impact of missing data on the primary analysis.

The SAS procedure MI will be used and the details of MI procedure will be stated in the dataset specification and TFL annotation document. If the data is monotone missing, a regression model will be used for imputation. Otherwise, the MCMC method will be used. All variables included

in the analysis model and values at month 3 for the corresponding endpoint will be included in the imputation model (Table 14.2.2.2a, Table 14.2.3.2a).

### 4.5 Analysis of Secondary Objectives

#### 4.5.1 Efficacy (Secondary)

Refer Section 4.4.2 for the analysis of secondary objectives.

#### 4.6 Exploratory Analysis

The exploratory efficacy variable is:

• Change from baseline in Insulin –like growth Factor-1 (IGF-1) at 3 and 6 months.

Summary statistics (n, mean, SD, SE, median, minimum and maximum) by product group and visit of the observed and change from baseline values will be provided (Table 14.2.19.1).

The change in baseline IGF-1 variable will be analyzed using the ANCOVA. The ANCOVA will have product group, age strata as fixed effects and the corresponding baseline value as covariate. Adjusted means, 95% confidence intervals, within product p-values for each product group difference, SE, 95% confidence interval of the difference and the between-product p-values based on the statistical model described above will be presented (Table 14.2.19.2). Statistical tests to compare treatments will be two-sided and will employ a level of significance of  $\alpha = 0.05$ .

Assumptions of normality and homogeneity of variances in the ANCOVA model will be evaluated after study un-blinding. If violations are observed then the following will be performed as a post-hoc sensitivity analysis and results will be compared with primary analysis results:

- 1. Suitable data transformations will be tried to achieve the assumptions.
- 2. If suitable transformations cannot be found, then the non-parametric Van Elteren tests will be performed adjusting for age strata for each endpoint.

To visually inspect the treatment effect on each of the secondary endpoints, plots across time (Baseline, Month 3 and Month 6) will be displayed with LSmeans and  $\pm$  SE bars which will be obtained from the ANCOVA analysis.. The plot will display a different symbol line for each treatment group (Figure 14.2.19.1).

Missing data will be handled as described in Section 4.4.3.

Seven day dietary intake assessment is conducted at baseline and at month 6.

GlaxoSmithKline Consumer Healthcare 

Observed values at each visit (baseline and month 6) and change from baseline at month 6 will be summarized descriptively (n, mean, standard deviation, median, minimum, and maximum) by product group (Table 14.2.20.1).

Seven day dietary intake assessments will be listed in Listing 16.2.6.21.

#### 4.6.1 Dietary Intake Assessment Post hoc Analyses

A post hoc ANCOVA analysis will be performed at Month 6 for each dietary intake parameter. The ANCOVA model will include the change in baseline dietary intake parameter as response variable and will have product group as fixed effects and the corresponding baseline values for each parameter as covariate. Adjusted means, 95% confidence intervals (CIs), within product p-values for each product group, product group difference, SE, 95% confidence interval of the difference and the between-product p-values based on the statistical model described above will also be presented (Table 14.2.20.2). Statistical tests to compare treatments will be two-sided and will employ a level of significance of  $\alpha = 0.05$ .

#### 4.6.2 Further Post hoc Analysis

This post hoc analysis will be performed on urine CTX-1 over creatinine ratio (CTX1CR). The efficacy variable is as follows:

• Change from baseline in CTX1CR after 3 and 6 months of treatment.

Summary statistics (n, mean, SD, SE, median, minimum and maximum) by product group and visit of the observed and change from baseline values will be provided for CTX1CR (Table 14.2.21.1).

The CTX1CR data will be provided in Listing 16.2.6.22.

The change from baseline in CTX1CR will be analysed using ANCOVA. The ANCOVA model will have product group, age strata as fixed effects and the corresponding baseline value as a covariate. Adjusted means, 95% confidence intervals, within product p-values for each product group, product group difference, SE, 95% confidence interval of the difference and the between-product p-values based on the statistical model described above will also be presented (Table 14.2.21.2). Statistical tests to compare treatments will be two-sided and will employ a level of significance of  $\alpha = 0.05$ .

Assumptions of normality and homogeneity of variances in the ANCOVA model will be evaluated. If violations are observed then the following will be performed as a post-hoc sensitivity analysis:

- 1. Suitable data transformations will be tried to achieve the assumptions.
- 2. If suitable transformations cannot be found, then the non-parametric Van Elteren tests will be performed adjusting for age strata for each endpoint.

GlaxoSmithKline Consumer Healthcare Confidential


### 4.7 Analysis of Safety

#### 4.7.1 Adverse Events and Serious Adverse Events

Adverse events (AE) recorded during the study will be mapped to a system organ class (SOC) and preferred term (PT) using the current medical dictionary for regulatory activities (MedDRA).

Treatment emergent adverse events (TEAEs) are defined as new AEs that occur on or after the date/time of the first administration of study product.

The following summary tables and listings will be presented by product group for safety population:

- Table of TEAEs by System Organ Class and Preferred Term (Table 14.3.1.1)
- Table of TEAEs related to study product by System Organ Class and Preferred Term (Table 14.3.1.2)
- Table of TEAEs by System Organ Class, Preferred Term and Severity (Table 14.3.1.3)
- Listing of all AEs (including all subjects: Listing 16.2.7.1.1 for all randomized subjects; Listing 16.2.7.1.2 for non-randomized subjects)
- Listing of death occurring during treatment (if any) will be listed by treatment, including the date and study day of death, and the principal cause of death (Listing 14.3.2.1)
- Listing of non-fatal serious adverse events (Listing 14.3.2.2)
- Listing of TEAEs leading to withdrawal (Listing 14.3.2.3)

#### 4.7.2 Laboratory Tests

Laboratory and biomarker results at screening, baseline, and each follow-up visit until end of the study visit will be presented in shift tables (Tables 14.3.5.3 - 14.3.5.12).

\* The tests are named according to the protocol. This naming convention of the parameters will be used for generating the outputs also.

Laboratory parameters for which reference ranges will be available will then be categorised with respect to reference ranges as: High, Low, Normal and Missing. The shift will be calculated with respect to reference ranges from baseline for the subsequent visits.

The reference ranges will not be available for the following laboratory tests –

Serum Cross-Linked C-Telopeptide of Type 1 Collagen, Ratio of Carboxylated to Under-Carboxylated Osteocalcin, Urinary C-Telopeptide of Type 1 Collagen, Serum Vitamin D (using 25-OH D3), Urinary Calcium/Creatinine Ratio and Serum Folate.

Laboratory normal ranges will be listed in Listing 16.2.6.20 and all laboratory test results will be listed in Listings 16.2.6.1 - 16.2.6.19.

#### 4.7.3 Vital Signs

Vital signs (systolic and diastolic blood pressure (mmHg), heart rate (beats/min), and oral body temperature (°F)) will be collected at screening, baseline, and each follow-up visit until end of the study visit.

Observed values at each visit and change from baseline at each post-baseline visit will be summarized on the safety population descriptively (n, mean, standard deviation, median, minimum, and maximum) by product group (Table 14.3.5.1).

All vital signs will listed in Listing 16.2.9.1.

#### 4.7.4 Findings on Physical Examination

The findings on the physical examination performed at screening, baseline, and each follow-up visit until end of the study visit will be listed (Listing 16.2.9.2).

#### 4.7.5 Other Safety Variables

Hemoglobin (g/dL) collected at screening, baseline, and each follow-up visit until end of the study visit will be summarized descriptively for all subjects in safety population.

Observed values at each visit and change from baseline at each post-baseline visit will be summarized descriptively (n, mean, standard deviation, median, minimum, and maximum) by product group (Table 14.3.5.2). Baseline will be defined as the last measurement before the first dose of study product; change will be defined as the post-baseline value minus the baseline value.

Hemoglobin measurements will be listed in Listing 16.2.9.3.

#### 4.8 Analysis of Other Variables

Not applicable.

#### 4.8.1 Quality of Life

Not applicable.


#### 4.8.2 Patch Adhesion Performance

Not applicable.

## 5 Changes to the Protocol Defined Statistical Analysis Plan

Any changes from the originally planned statistical analysis specified in the protocol (Dated: 31/JUL/2017) are outlined in Table .

Table 2 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis section | Statistical Analysis Plan | Rationale for Changes |
| Section 9.2.1 | Section 4.1.3 | PP population definition is clarified<br>and elaborated. Partial (in case of<br>non-compliance in any particular<br>visits) and full exclusion are<br>defined. |
| <ul><li>Section 9.3.2</li><li>Section 9.3.3</li></ul> | <ul> <li>Section 4.4.1.2</li> <li>Section 4.5.1</li> <li>Section 4.6</li> </ul> | <ul> <li>ANCOVA model for the primary, secondary and exploratory analysis has been updated. Age strata have been added as a fixed effect in the model to account for the baseline stratification.</li> <li>Also, 95% CI is being updated with 97.5% CI since the significance level for the primary analysis is 0.025.</li> </ul> |

#### RAP Addendum 1

This RAP addendum v1.0 provides details of the additional analyses requested from the analyses described in the Statistical Reporting and Analysis Plan Amendment 1.The additional post-hoc analyses were identified at the non-topline TFL review stage, and hence was after un-blinding but prior to development of the CSR. The additional post-hoc analyses will be discussed in the CSR.

Sections 4.3.1.1, 4.4.1, 4.4.1.4, 4.4.2, and 4.6.1 were added in the RAP addendum describing the additional post-hoc analyses. The sections below provide a summary of this with the justification for the request.

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis | Statistical Analysis Plan Rationale for Changes | |
| section | _ | _ |

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis | Statistical Analysis Plan | Rationale for Changes |
| section | | |
| Section 5.5 | Section 4.3.1 | <ul> <li>Added Section 4.3.1.1 which details a study product compliance summary by categories 0-3 months and 3-6 months.</li> <li>This is to assess if the difference in compliance between the time points could be linked to the difference in primary parameter results between Month 3 and Month 6.</li> </ul> |
| Section 9.3.2 | Section 4.4.1 | Added a statistical model for the log-transformed data of s-CTX1 to support sensitivity analysis. |
| Section 9.3.2 | • Section 4.4.1.2 | Added Section 4.4.1.4 which details a subgroup ANCOVA analysis on s-CTX1 change from baseline by age strata at Month 3 and Month 6. This is to asses if age has an impact on the treatment effect. |
| • | • | • |
| Section 6.10 | Section 4.6 | Added Section 4.6.1 which details<br>an ANCOVA analysis on the<br>change from baseline of each<br>dietary intake parameter<br>assessment. This is to assess if<br>significant changes in dietary<br>intake can be linked to the change<br>in primary endpoint at Month 6. |

#### • RAP Addendum 2

This RAP addendum v2.0 provides details of the further post hoc analyses requested from the analysis described in the Statistical Reporting and Analysis Plan Addendum 1. This further post hoc analyses were identified after submission of all final TFLs, and hence after un-blinding. The further post-hoc analysis will be discussed in the CSR.

The section below provides a summary of the further post hoc analysis with the justification for the request.

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis | Statistical Analysis Plan | Rationale for Changes |
| section | | |
| Not Applicable | • Section 4.6.2 | Added Section 4.6.2 which details<br>ANCOVA analysis of new variable<br>urine CTX-1 over creatinine ratio.<br>The rationale of this new analysis<br>is to account for the impact of<br>dilution and kidney function on<br>urinary values, and to explore<br>further the difference between<br>urine and serum CTX-1 results. |

## **Attachment 1: List of Data Displays**



## 6 Template for Tables, Figures and Listings

This is a guideline which will give the guidance of product labels that will be used for the table header and in the figures, listings and in the footnotes.

The product labels for the column headings will be as follow:

- Test Product
- Reference Product

The product comparison will be:

• Test Product vs Reference Product

The below footnotes will be displayed on each output

- Test Product: Cereal based fortified beverage (Proprietary food)
- Reference Product: Low protein non fortified isocaloric beverage

Final Statistical Reporting and Analysis Plan Addendum Version 2.0 23-July-2018

Protocol 207192 Program Run Date: DDMMMYYYY

Table 14.1.1 Subject Disposition All Screened Subjects

Study Population: All Screened Subjects (N=xxx)

| | Test Product | Reference Product | Overall |
|---|---|---|---|
| | n (%) | n (%) | n (%) |
| TOTAL SUBJECTS SCREENED | | | xxx |
| SUBJECTS NOT RANDOMIZED DID NOT MEET STUDY CRITERIA | | | xxx (xx.x) |
| ADVERSE EVENT | | | xxx (xx.x)<br>xxx (xx.x) |
| SUBJECTS RANDOMIZED | XXX | XXX | XXX |
| COMPLETED STUDY DID NOT COMPLETE STUDY | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| DID NOT MEET STUDY CRITERIA | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| ADVERSE EVENT | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| LOST TO FOLLOW-UP | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| PROTOCOL VIOLATION | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| WITHDRAWAL OF CONSENT | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| OTHER | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| SAFETY POPULATION | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| ITT POPULATION | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| PP POPULATION | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Percentages for not randomized category are based on number of screened subjects; percentages for randomized category are based on number of randomized subjects.

Page x of y

Program: xxxxxx.sas Source: Filename


Protocol 207192 Program Run Date: DDMMYYYY

# Table 14.1.2 Incidence of Major Protocol Deviations Randomized Population

Study Population: Randomized (N=xxx)

| | Test Product | Reference Product | Overall |
|---|---|---|---|
| | n (%) | n (%) | n (%) |
| SUBJECTS WITH AT LEAST ONE MAJOR PROTOCOL DEVIATION | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| MAJOR PROTOCOL DEVIATIONS NOT LEADING TO EXCLUSION FROM PP | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| DEVIATION REASON 1 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| MAJOR PROTOCOL DEVIATIONS LEADING TO EXCLUSION FROM PP | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| All VISITS | | | |
| DEVIATION REASON 1 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| VISIT Y | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| DEVIATION REASON 1 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

**Programming Note:** This table will list all major protocol deviations as defined in the population definition document.


Protocol: 207192 Program Run Date: DDMMMYYYY

# Table 14.1.4.1 Demographic and Baseline Characteristics Safety Population

Study Population: Safety Population (N=XXX)

| paration. Survey reparation (17-7000) | Test Product | Reference Product | Overall |
|---|---|---|---|
| | (N = xxx) | (N = xxx) | (N = xxx) |
| RACE n (%) | | | |
| AFRICAN AMERICAN/AFRICAN HERITAGE | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| AMERICAN INDIAN OR ALASKAN NATIVE | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| AGE (YEARS) | | | |
| n | xx | xx | xx |
| MEAN | XX.X | xx.x | xx.x |
| AGE GROUP n (%) | | | |
| ≥ 25 - < 35 YEARS | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| ≥ 35 - ≤ 45 YEARS | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| SEX n (%) | | | |
| FEMALE | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| HEIGHT (cm) | | | |
| n | XX | xx | xx |
| MEAN | xxx.xx | XXX.XX | xxx.xx |
| WEIGHT (kg) | | | |
| n | xx | xx | xx |
| MEAN | XXX.XX | xxx.xx | xxx.xx |


| DDY MASS INDEX (kg/m²) | | | |
|------------------------|--------|--------|--------|
| n | xx | xx | xx |
| MEAN | XXX.XX | xxx.xx | xxx.xx |

**Programming Note:** For continuous variables the summary statistics: n, Mean, SD, Median, Minimum and Maximum will be displayed. Similar table will be displayed for ITT population.


Protocol 207192 Program Run Date: DDMMMYYYY

Table 14.2.1.1 Study Product Compliance Intent-to-Treat Population

Study Population: Intent-to-Treat Population (N = xxx) Statistics Test Product Reference Product (N = xxx)(N = xxx)TOTAL NUMBER OF SACHETS DISPENSED XX XX MEAN x.xxx x.xxx SD x.xxxx x.xxxx MEDIAN X.XXX x.xxx MINIMUM X.XX X.XX MAXIMUM x.xx x.xx TOTAL NUMBER OF SACHETS CONSUMED XX XX MEAN x.xxx x.xxx SD x.xxxx X.XXXX MEDIAN X.XXX x.xxx MINIMUM X.XX X.XX MAXIMUM X.XX X.XX TOTAL NUMBER OF SACHETS RETURNED XX XX MEAN x.xxx x.xxx SD x.xxxx x.xxxx MEDIAN x.xxx x.xxx MINIMUM X.XX X.XX MAXIMUM X.XX X.XX COMPLIANCE XX XX MEAN X.XXX x.xxx x.xxxx X.XXXX MEDIAN x.xxx x.xxx MINIMUM x.xx x.xx MAXIMUM x.xx X.XX


| | Statistics | Test Product<br>(N = xxx) | Reference Product<br>(N = xxx) |
|---|---|---|---|
| NUMBER OF SUBJECTS COMPLIANT NUMBER OF SUBJECTS NON-COMPLIANT | n (%) | xxx (xx.x) | xxx (xx.x) |
| | n (%) | xxx (xx.x) | xxx (xx.x) |

Percentage is based on number of subjects in each product group.

Subject would be considered non-compliant if the subject consumes less than 80% of the total amount of recommended dose.

Compliance = (actual total number of sachets consumed/expected total number of sachets consumed)\*100 where,

actual number of sachets consumed = (number of sachets dispensed – number of sachets unconsumed returned)

Program: xxxxxx.sas Source: Filename

Page x of y

Protocol 207192 Program Run Date: DDMMMYYYY

#### Table 14.2.1.1a Study Product Compliance by Time Categories Intent-to-Treat Population

Study Population: Intent-to-Treat Population (N = xxx)

Time Category: 0-3 Months

| | Statistics | Test Product | Reference Product |
|---|---|---|---|
| | | (N = xxx) | (N = xxx) |
| TOTAL NUMBER OF SACHETS DISPENSED | | | |
| TO THE HOLDER OF STRONE IS DIST ENGES | n | XX | XX |
| | MEAN | x.xxx | x.xxx |
| | SD | X.XXXX | x.xxxx |
| | MEDIAN | x.xxx | x.xxx |
| | MINIMUM | X.XX | X.XX |
| | MAXIMUM | x.xx | x.xx |
| TOTAL NUMBER OF SACHETS CONSUMED | n | XX | xx |
| | MEAN | x.xxx | x.xxx |
| | SD | x.xxxx | x.xxxx |
| | MEDIAN | x.xxx | x.xxx |
| | MINIMUM | x.xx | x.xx |
| | MAXIMUM | x.xx | x.xx |
| TOTAL NUMBER OF SACHETS RETURNED | n | XX | XX |
| | MEAN | X.XXX | x.xxx |
| | SD | X.XXXX | X.XXXX |
| | MEDIAN | x.xxx | x.xxx |
| | MINIMUM | X.XX | X.XX |
| | MAXIMUM | x.xx | x.xx |
| COMPLIANCE | n | xx | XX |
| | MEAN | x.xxx | x.xxx |
| | SD | x.xxxx | x.xxxx |
| | MEDIAN | x.xxx | x.xxx |
| | MINIMUM | X.XX | X.XX |


| | Statistics | Test Product<br>(N = xxx) | Reference Product<br>(N = xxx) |
|---|---|---|---|
| | MAXIMUM | X.XX | X.XX |
| NUMBER OF SUBJECTS COMPLIANT NUMBER OF SUBJECTS NON-COMPLIANT | n (%)<br>n (%) | xxx (xx.x)<br>xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x) |

Percentage is based on number of subjects in each product group.

Subject would be considered non-compliant if the subject consumes less than 80% of the total amount of recommended dose.

Compliance = (actual total number of sachets consumed/expected total number of sachets consumed)\*100 where,

actual number of sachets consumed = (number of sachets dispensed – number of sachets unconsumed returned)

Page x of y

Program: xxxxxx.sas Source: Filename


Protocol 207192 Program Run Date: DDMMMYYYY

Table 14.2.2.1
Summary of Serum Cross Linking C-Telopeptide of Type 1 Collagen (Unit)
Intent-to-Treat Population

Study Population: Intent-to-Treat Population (N = xxx)

| Visit | Statistics | | roduct<br>xxx) | | ence Product<br>N = xxx) | Overall<br>(N = xxx) | |
|---|---|---|---|---|---|---|---|
| | | Observed Value | Change from Baseline | Observed Value | Change from Baseline | Observed Value | Change from Baseline |
| BASELINE | n | xxx | | xxx | | xxx | |
| | MEAN | xx.xx | | XX.XX | | XX.XX | |
| | SD | xx.xxx | | XX.XXX | | XX.XXX | |
| | SE | x.xx | | X.XX | | X.XX | |
| | MEDIAN | x.xx | | X.XX | | X.XX | |
| | MINIMUM | xx.x | | XX.X | | XX.X | |
| | MAXIMUM | XX.X | | xx.x | | XX.X | |
| MONTH 3 | n | xxx | XXX | xxx | XXX | | |
| | MEAN | xx.xx | xx.xx | xx.xx | xx.xx | | |
| | SD | xx.xxx | xx.xxx | XX.XXX | xx.xxx | | |
| | SE | x.xx | x.xx | X.XX | x.xx | | |
| | MEDIAN | x.xx | x.xx | X.XX | x.xx | | |
| | MINIMUM | xx.x | xx.x | XX.X | xx.x | | |
| | MAXIMUM | XX.X | XX.X | xx.x | XX.X | | |
| MONTH 6 | n | xxx | XXX | xxx | XXX | | |
| | MEAN | xx.xx | xx.xx | xx.xx | xx.xx | | |
| | SD | xx.xxx | xx.xxx | xx.xxx | xx.xxx | | |
| | SE | X.XX | x.xx | x.xx | x.xx | | |
| | MEDIAN | x.xx | x.xx | x.xx | x.xx | | |
| | MINIMUM | xx.x | xx.x | xx.x | xx.x | | |
| | MAXIMUM | xx.x | xx.x | XX.X | xx.x | | |


**Programming Note:** Similar table will be generated for all other primary, secondary and exploratory variables. Overall column will be displayed only for the Baseline visits.

Protocol 207192 Program Run Date: DDMMMYYYY

# Table 14.2.2.1a Summary of Serum Cross Linking C-Telopeptide of Type 1 Collagen (Unit) by Age Strata Intent-to-Treat Population

Study Population: Intent-to-Treat Population (N = xxx)

Strata 1: 25 -<35 years

| Visit | Statistics | | roduct<br>xxx) | | ence Product<br>N = xxx) | Overall<br>(N = xxx) | |
|---|---|---|---|---|---|---|---|
| | | Observed Value | Change from Baseline | Observed Value | Change from Baseline | Observed Value | Change from Baseline |
| BASELINE | n | xxx | | xxx | | xxx | |
| | MEAN | xx.xx | | xx.xx | | XX.XX | |
| | SD | xx.xxx | | XX.XXX | | XX.XXX | |
| | SE | x.xx | | X.XX | | X.XX | |
| | MEDIAN | x.xx | | X.XX | | X.XX | |
| | MINIMUM | xx.x | | xx.x | | XX.X | |
| | MAXIMUM | XX.X | | XX.X | | XX.X | |
| MONTH 3 | n | XXX | XXX | xxx | XXX | | |
| | MEAN | xx.xx | xx.xx | xx.xx | xx.xx | | |
| | SD | xx.xxx | xx.xxx | xx.xxx | xx.xxx | | |
| | SE | x.xx | x.xx | x.xx | x.xx | | |
| | MEDIAN | x.xx | x.xx | X.XX | x.xx | | |
| | MINIMUM | xx.x | xx.x | XX.X | xx.x | | |
| | MAXIMUM | XX.X | XX.X | xx.x | XX.X | | |
| MONTH 6 | n | XXX | XXX | xxx | XXX | | |
| | MEAN | xx.xx | xx.xx | xx.xx | xx.xx | | |
| | SD | xx.xxx | xx.xxx | xx.xxx | xx.xxx | | |
| | SE | x.xx | x.xx | x.xx | x.xx | | |
| | MEDIAN | x.xx | x.xx | x.xx | x.xx | | |
| | MINIMUM | XX.X | xx.x | XX.X | xx.x | | |
| | MAXIMUM | xx.x | xx.x | XX.X | xx.x | | |


| - | | | | |
|-------|------------|--------------|-------------------|-----------|
| Visit | Statistics | Test Product | Reference Product | Overall |
| | | (N = xxx) | (N = xxx) | (N = xxx) |


Protocol 207192 Program Run Date: DDMMMYYYY

# Table 14.2.2.2 Statistical Analysis of Serum Cross Linking C-Telopeptide of Type 1 Collagen (Unit) Change from Baseline Intent-to-Treat Population

Study Population: Intent-to-Treat Population (N = xxx)

| Vicit | Dradust Craun | | | | | Comparison with Reference Product | | | |
|---|---|---|---|---|---|---|---|---|---|
| Visit | Product Group | N | Adjusted Mean | SE | 95% CI | P-Value | Difference (SE) | 97.5% CI | P-Value |
| MONTH 3 | TEST PRODUCT<br>REFERENCE PRODUCT | xxx<br>xxx | xx.xx<br>xx.xx | xx.xxx<br>xx.xxx | xx.xx, xx.xx<br>xx.xx, xx.xx | 0.xxxx<br>0.xxxx | xx.xx (xx.xxx) | xx.xx, xx.xx | 0.xxxx |
| MONTH 6* | TEST PRODUCT<br>REFERENCE PRODUCT | xxx<br>xxx | XX.XX<br>XX.XX | xx.xxx<br>xx.xxx | xx.xx, xx.xx<br>xx.xx, xx.xx | 0.xxxx<br>0.xxxx | xx.xx (xx.xxx) | xx.xx, xx.xx | 0.xxxx |

<sup>\*</sup> one of the co-primary efficacy endpoints.

Program: xxxxxx.sas

Analysis was performed using ANCOVA model with product group, age strata as fixed effects and the corresponding baseline value as covariate. Difference is test product minus reference product such that a negative difference favors the test product.

Source: Filename

Page x of y

**Programming Note:** Similar table will be generated for all primary endpoints. Direction of the difference should be with respect to the parameter which will be analyzed and should be checked with Clinical Research and Statistician for finalization. For month 3, alpha value will be used 0.05 and the confidence intervals for within and between comparisons will be of 95%. For month 6, alpha will be used 0.05 for the within and for between product group comparisons alpha will be 0.025 and the confidence interval will be 97.5%.

Show month 3 values in page 1 and month 6 values in page 2.


Protocol 207192 Program Run Date: DDMMMYYYY

# Table 14.2.2.2a Statistical Analysis of Serum Cross Linking C-Telopeptide of Type 1 Collagen (Unit) Change from Baseline using Imputed Missing Data Safety Population

Study Population: Intent-to-Treat Population (N = xxx)

| Visit | Draduat Craus | | | | | | Comparis | son with Reference Proc | luct |
|---|---|---|---|---|---|---|---|---|---|
| VISIL | Product Group | N | Adjusted Mean | SE | 95% CI | P-Value | Difference (SE) | 97.5% CI | P-Value |
| MONTH 6* | TEST PRODUCT<br>REFERENCE PRODUCT | xxx<br>xxx | XX.XX<br>XX.XX | xx.xxx<br>xx.xxx | xx.xx, xx.xx<br>xx.xx, xx.xx | 0.xxxx<br>0.xxxx | xx.xx (xx.xxx) | xx.xx, xx.xx | 0.xxxx |

<sup>\*</sup>one of the co-primary efficacy endpoints.

To impute the monotone missing pattern data a regression model method will be applied with following effects; product group, age strata and the corresponding baseline and Month 3 data will be used.

Analysis was performed using ANCOVA model with product group, age strata as fixed effects and the corresponding baseline value as covariate. Difference is test product minus reference product such that a negative difference favors the test product.

Page x of y

Program: xxxxxx.sas Source: Filename

**Programming Note:** Similar table will be generated for all primary endpoints using imputed missing data. Direction of the difference should be with respect to the parameter which will be analyzed and should be checked with Clinical Research and Statistician for finalization.

For month 3, alpha value will be used 0.05 and the confidence intervals for within and comparisons will be of 95%. For month 6, alpha will be used 0.05 for the within and for between product group comparisons alpha will be 0.025 and the confidence interval will be 97.5%. Show month 3 values in page 1 and month 6 values in page 2.


Protocol 207192 Program Run Date: DDMMMYYYY

## Table 14.2.2.2b Statistical Analysis of Serum Cross Linking C-Telopeptide of Type 1 Collagen (Unit) Change from Baseline by Age Strata Intent-to-Treat Population

Study Population: Intent-to-Treat Population (N = xxx)

Age Strata: 25-<35 years

| Visit | Product Group | | | | | | Compari | ison with Reference Pro | duct |
|---|---|---|---|---|---|---|---|---|---|
| VISIL | Product Group | N | Adjusted Mean | SE | 95% CI | P-Value | Difference (SE) | 97.5% CI | P-Value |
| MONTH 3 | TEST PRODUCT<br>REFERENCE PRODUCT | xxx<br>xxx | xx.xx<br>xx.xx | xx.xxx<br>xx.xxx | xx.xx, xx.xx<br>xx.xx, xx.xx | 0.xxxx<br>0.xxxx | xx.xx (xx.xxx) | xx.xx, xx.xx | 0.xxxx |
| MONTH 6* | TEST PRODUCT<br>REFERENCE PRODUCT | xxx<br>xxx | xx.xx<br>xx.xx | xx.xxx<br>xx.xxx | xx.xx, xx.xx<br>xx.xx, xx.xx | 0.xxxx<br>0.xxxx | xx.xx (xx.xxx) | xx.xx, xx.xx | 0.xxxx |

<sup>\*</sup> one of the co-primary efficacy endpoints.

Analysis was performed using ANCOVA model with product group, strata and product\*strata interaction as fixed effects and the corresponding baseline value as covariate. Difference is test product minus reference product such that a negative difference favors the test product.

Page x of y

Program: xxxxxx.sas Source: Filename

**Programming Note:** Similar table will be generated for all primary endpoints. Direction of the difference should be with respect to the parameter which will be analyzed and should be checked with Clinical Research and Statistician for finalization. For month 3 and month 6, alpha value will be used 0.05 and the confidence intervals for within and between comparisons will be of 95%.


Protocol 207192 Program Run Date: DDMMMYYYY

# Table 14.2.2.2c Statistical Analysis of Serum Cross Linking C-Telopeptide of Type 1 Collagen (Unit) using Log Transformed Data Intent-to-Treat Population

#### Study Population: Intent-to-Treat Population (N = xxx)

| | | | | | | | Comparison with Reference Product | | |
|---|---|---|---|---|---|---|---|---|---|
| Visit | Product Group | N | Geometric Mean | Geometric CV | 95% CI | P-Value | Geometric Mean Ratio<br>(CV) | 95% CI | P-Value |
| MONTH 3 | TEST PRODUCT<br>REFERENCE PRODUCT | xxx<br>xxx | xx.xx<br>xx.xx | xx.xxx<br>xx.xxx | xx.xx, xx.xx<br>xx.xx, xx.xx | 0.xxxx<br>0.xxxx | xx.xx (xx.xxx) | xx.xx, xx.xx | 0.xxxx |

Analysis was performed for log transformed data using ANCOVA model with product group, age strata as fixed effects and the corresponding log(baseline) value as covariate. Geometric mean ratio less than one favors the

Page x of y

Program: xxxxxx.sas

Source: Filename

#### **Programming Note:**

For Month 6 create a new page and use alpha as 0.025 and 97.5% CI. Geometric mean = exp (LSmean); Geometric CV = sqrt(exp(variance)-1); Geometric mean ratio =exp(difference); Lower CI = exp(LCL) and Upper CI = exp(UCL)


Protocol 207192 Program Run Date: DDMMMYYYY

# Table 14.2.4.2 Statistical Analysis of Urinary C-Telopeptide of Type 1 Collagen (Unit) Change from Baseline Intent-to-Treat Population

Study Population: Intent-to-Treat Population (N = xxx)

| Visit | Product Group | | | | | | Compar | ison with Reference Pro | duct |
|---|---|---|---|---|---|---|---|---|---|
| VISIL | Product Group | N | Adjusted Mean | SE | 95% CI | P-Value | Difference (SE) | 95% CI | P-Value |
| MONTH 3 | TEST PRODUCT<br>REFERENCE PRODUCT | xxx<br>xxx | xx.xx<br>xx.xx | xx.xxx<br>xx.xxx | xx.xx, xx.xx<br>xx.xx, xx.xx | 0.xxxx<br>0.xxxx | xx.xx (xx.xxx) | xx.xx, xx.xx | 0.xxxx |
| MONTH 6 | TEST PRODUCT<br>REFERENCE PRODUCT | xxx<br>xxx | xx.xx<br>xx.xx | xx.xxx<br>xx.xxx | xx.xx, xx.xx<br>xx.xx, xx.xx | 0.xxxx<br>0.xxxx | xx.xx (xx.xxx) | xx.xx, xx.xx | 0.xxxx |

Analysis was performed using ANCOVA model with product group, age strata as fixed effects and the corresponding baseline value as covariate. Difference is test product minus reference product such that a negative difference favors the test product.

Page x of y
Program: xxxxxx.sas Source: Filename

**Programming Note:** Similar table will be generated for all secondary and exploratory endpoints. Direction of the difference should be with respect to the parameter which will be analyzed and should be checked with Clinical Research and Statistician for finalization.


Protocol 207192 Program Run Date: DDMMMYYYY

# Table 14.2.9.2a Statistical Analysis of Calcium/Creatinine Ratio (unit) using Log Transformed Data Intent-to-Treat Population

Study Population: Intent-to-Treat Population (N = xxx)

| | | | | | | | | | | Comparison with Reference Product |
|---|---|---|---|---|---|---|---|---|---|---|
| Visit | Product Group | N | Geometric Mean | Geometric CV | 95% CI | P-Value | Geometric Mean Ratio | 95% CI | P-Value | |
| | | | | | | | (CV) | | | |
| MONTH 3 | TEST PRODUCT | xxx | xx.xx | xx.xxx | xx.xx, xx.xx | 0.xxxx | xx.xx (xx.xxx) | xx.xx, xx.xx | 0.xxxx | |
| | REFERENCE PRODUCT | XXX | xx.xx | xx.xxx | xx.xx, xx.xx | 0.xxxx | | | | |
| MONTH 6 | TEST PRODUCT | xxx | xx.xx | xx.xxx | xx.xx, xx.xx | 0.xxxx | xx.xx (xx.xxx) | xx.xx, xx.xx | 0.xxxx | |
| | REFERENCE PRODUCT | xxx | xx.xx | xx.xxx | xx.xx, xx.xx | 0.xxxx | | | | |

Analysis was performed for log transformed data using ANCOVA model with product group, age strata as fixed effects and the corresponding log(baseline) value as covariate. Geometric mean ratio less than one favors the test product.

Page x of y
Program: xxxxxxx.sas Source: Filename

#### **Programming Note:**

Geometric mean = exp (LSmean); Geometric CV = sqrt(exp(variance)-1); Geometric mean ratio =exp(difference); Lower CI = exp(LCL) and Upper CI = exp(UCL)


Protocol 207192 Program Run Date: DDMMMYYYY

#### Table 14.2.20.1 Summary of Seven Day Dietary Intake Assessment ITT Population

Study Population: ITT Population (N = xxx)

| Parameter (Unit) | Visit | Statistics | | Product<br>= xxx) | Reference P<br>(N = xx: | | Overall<br>(N = xxx) |
|---|---|---|---|---|---|---|---|
| | | | Observed Value | Change from Baseline | Observed Value | Change from<br>Baseline | Observed Value |
| TOTAL ENERGY INTAKE (KCAL) | BASELINE | n | XXX | | XXX | | xxx |
| | | MEAN | xxx.x | | XXX.X | | xxx.x |
| | | SD | xxx.xx | | XXX.XX | | xxx.xx |
| | | MEDIAN | xxx.x | | XXX.X | | xxx.x |
| | | MINIMUM | xxx | | XXX | | xxx |
| | | MAXIMUM | Xxx | | Xxx | | Xxx |
| | MONTH 6 (VISIT 6) | n | XXX | xxx | xxx | xxx | |
| | | MEAN | xxx.x | xxx.x | xxx.x | xxx.x | |
| | | SD | xxx.xx | xxx.xx | xxx.xx | xxx.xx | |
| | | MEDIAN | xxx.x | xxx.x | xxx.x | xxx.x | |
| | | MINIMUM | xxx | xxx | XXX | XXX | |
| | | MAXIMUM | Xxx | Xxx | Xxx | Xxx | |

**Programming Note:** This table will continue for all parameters for dietary intake assessment [Total Energy intake (Kcal), Total Carbohydrate intake (gm), Total Fat intake (gm), Avergare Calcium intake (mg), Average protein intake (g), Average Vitamin D intake (mcg), Average Vitamin B6 intake (mg), Average Vitamin B12 intake (mg), Average Phosphorous intake (mg), Average Folic Acid intake (mcg), Average Zinc intake (mg), and Average Selenium intake (mcg)]. Display overall only for the baseline visit.


Protocol 207192 Program Run Date: DDMMMYYYY

#### Table 14.2.20.2 Statistical Analysis of Dietary Intake) Change from Baseline by Parameter Intent-to-Treat Population

Study Population: Intent-to-Treat Population (N = xxx)

Parameter: Total Energy (Kcal)

| Visit | Due doet Cuerre | | | | | | Comparison with Reference Product | | |
|---|---|---|---|---|---|---|---|---|---|
| | Product Group | N | Adjusted Mean | SE | 95% CI | P-Value | Difference (SE) | 95% CI | P-Value |
| MONTH 6 | TEST PRODUCT | XXX | xx.xx | xx.xxx | xx.xx, xx.xx | 0.xxxx | xx.xx (xx.xxx) | xx.xx, xx.xx | 0.xxxx |
| | REFERENCE PRODUCT | XXX | XX.XX | xx.xxx | xx.xx, xx.xx | 0.xxxx | | | |

Analysis was performed using ANCOVA model with product group, age strata as fixed effects and the corresponding baseline value as covariate. Difference is test product minus reference product such that a positive difference favors the test product.

Program: xxxxxx.sas Source: Filename Page x of y

**Programming Note:** This table will continue for all parameters for dietary intake assessment [Total Energy intake (Kcal), Total Carbohydrate intake (gm), Total Fat intake (gm), Avergare Calcium intake (mg), Average protein intake (g), Average Vitamin D intake (mcg), Average Vitamin B6 intake (mg), Average Vitamin B12 intake (mg), Average Phosphorous intake (mg), Average Folic Acid intake (mcg), Average Zinc intake (mg), and Average Selenium intake (mcg)].


Protocol 207192 Program Run Date: DDMMYYYY

Table 14.3.1.1

Treatment Emergent Adverse Event by System Organ Class and Preferred Term Safety Population

| Study Population: Safety Population (N=xxx) |
|---------------------------------------------|
|---------------------------------------------|

| System Organ Class<br>Preferred Term | Test Pro<br>(N = x) | | Reference<br>(N = ) | | Overall<br>(N = xxx) | |
|---|---|---|---|---|---|---|
| | n (%) | nAE | n (%) | nAE | n (%) | nAE |
| NUMBER OF SUBJECTS WITH AT LEAST ONE AE | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx |
| NUMBER OF SUBJECTS WITH NO AE | xx (xx.x) | | xx (xx.x) | | xx (xx.x) | |
| SOC 1 | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx |
| PT 1 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| PT 2 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| SOC 2 | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx |
| PT 1 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | xx |
| PT 2 | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx |

n (%) = Number (percent) of subjects; nAE = Number of adverse events.

Program: xxxxxx.sas Source: Filename Page x of y

**Programming Note:** Similar table will be generated for treatment related adverse events.


Protocol 207192 Program Run Date: DDMMYYYY

Table 14.3.1.3

Treatment Emergent Adverse Event by System Organ Class, Preferred Term and Severity
Safety Population

Study Population: Safety Population (N=xxx)

| System Organ Class<br>Preferred Term | Test Product<br>(N = xxx) | | | | | Reference Product<br>(N = xxx) | | | | Overall<br>(N = xxx) | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Mile | d | Mode | rate | Seve | ere | Milo | ł | Mode | rate | Seve | re | Mile | d | Moder | ate | Sever | re |
| | n (%) | nAE | n (%) | nAE | n (%) | nAE | n (%) | nAE | n (%) | nAE | n (%) | nAE | n (%) | nAE | n (%) | nAE | n (%) | nAE |
| SOC 1<br>PT 1<br>PT 2 | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx<br>xx<br>xx | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx<br>xx<br>xx | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx<br>xx<br>xx | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx<br>xx<br>xx | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx<br>xx<br>xx | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx<br>xx<br>xx | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx<br>xx<br>xx | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx<br>xx<br>xx | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx<br>xx<br>xx |

n (%) = Number (percent) of subjects; nAE = Number of adverse events.

Program: xxxxxx.sas Source: Filename Page x of y

Fortified HFD 207192


Protocol 207192 Program Run Date: DDMMMYYYY

Table 14.3.5.1 Summary of Vital Signs Safety Population

Study Population: Safety Population (N = xxx) Vital Sign: <Parameter Name (Unit)>

| Visit | Statistics | | roduct<br>xxx) | | ence Product<br>N = xxx) | Overall (N = xxx) |
|---|---|---|---|---|---|---|
| | | Observed Value | Change from Baseline | Observed Value | Change from Baseline | Observed Value |
| SCREENING | n | xxx | | XXX | | xxx |
| | MEAN | xxx.x | | XXX.X | | XXX.X |
| | SD | xxx.xx | | XXX.XX | | XXX.XX |
| | MEDIAN | xxx.x | | XXX.X | | XXX.X |
| | MINIMUM | XXX | | XXX | | XXX |
| | MAXIMUM | Xxx | | Xxx | | Xxx |
| BASELINE | n | XXX | | xxx | | xxx |
| S/ (SELINE | MEAN | XXX.X | | XXX.X | | XXX.X |
| | SD | xxx.xx | | XXX.XX | | XXX.XX |
| | MEDIAN | xxx.x | | XXX.X | | XXX.X |
| | MINIMUM | xxx | | XXX | | xxx |
| | MAXIMUM | Xxx | | Xxx | | Xxx |
| /ISIT 3 | n | xxx | XXX | xxx | XXX | |
| | MEAN | XXX.X | xxx.x | XXX.X | xxx.x | |
| | SD | xxx.xx | xxx.xx | XXX.XX | xxx.xx | |
| | MEDIAN | xxx.x | xxx.x | xxx.x | xxx.x | |
| | MINIMUM | xxx | xxx | XXX | xxx | |
| | MAXIMUM | Xxx | Xxx | Xxx | Xxx | |

**Programming Note:** This table will continue for all other scheduled visits and for all vital signs [Systolic blood pressure (mmHg), Diastolic blood pressure (mmHg), Heat rate (beats/min) and Oral body temperature (°F)]. Display overall only for the baseline visit.


Protocol 207192 Program Run Date: DDMMMYYYY

# Table 14.3.5.3 Shift Table for Serum N-Terminal Telopeptide of Type 1 Collagen (unit) Safety Population

Study Population: Safety Population (N = xxx)
Reference range: <xx-xx>,

| | | | F | | Re | ference Prod | uct | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Baseline | | | | | Baseline | | |
| Visit | Result | Low<br>n (%) | Normal<br>n (%) | High<br>n (%) | Missing<br>n (%) | Total<br>n (%) | Low<br>n (%) | Normal<br>n (%) | High<br>n (%) | Missing<br>n (%) | Total<br>n (%) |
| Month 3 | Low | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX<br>(XX.X) |
| | Normal<br>High<br>Missing<br>Total | | | | | | | | | | |
| Month 6 | Low | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX<br>(XX.X) |
| | Normal<br>High<br>Missing<br>Total | | | | | | | | | | |

**Programming Note:** This table will continue for all other scheduled visits and laboratory parameters


Protocol 207192 Program Run Date: DDMMYYYY

# Listing 16.1.7 Randomization Information All Randomized Subjects

| Subject Number | Age/Race [1] | Strata | Randomization Number | Product Group | Date of Randomization |
|---|---|---|---|---|---|
| XXXXXX | XX/A1 | Stratum 1: Age ≥ 25 - 35 years | xxxxxx | | DDMMMYYYY |

---

[1] Age in years; Race: A1 = African American/African Heritage, A2 = American Indian Or Alaskan Native, A3 = Asian-Central/South Asian Heritage, A4 = Asian-East Asian Heritage, A5 = Asian-Japanese Heritage, A6 = Asian-South East Asian Heritage, N = Native Hawaiian Or Other Pacific Islander, W1 = White-Arabic/North African Heritage, W2 = White - White/Caucasian/European Heritage, MT = Multiple.

The block size of X was used for this randomization.

Page x of y

Program: xxxxxx.sas

Source: Filename

**Programming Note:** Block size information will be added after un-blinding of the treatment code.


Protocol 207192 Program Run Date: DDMMYYYY

Listing 16.2.1.1.1 Subject Disposition All Randomized Subjects

Study Population: All Randomized Subjects(N=xx)

| Pro | duct | Group | · xxxx | (XX |
|-----|------|-------|--------|-----|

| r roudet Group | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Age/Race [1] | Screening Date | Study Product Start<br>Date and Time | Last Study Product Administration Date and Time | Date of Completion<br>or Withdrawal | Duration in the<br>Study (days) [2] | Completed the<br>Study | Primary Reason for<br>Withdrawal | Further Details [3] |
| xxxxxx | XX/A1 | DDMMMYYYY | DDMMMYYYY:HH:M<br>M | DDMMMYYYY:HH:MM | DDMMMYYYY | xxx | Yes | | |
| XXXXXX | XX/A6 | DDMMMYYYY | DDMMMYYYY:HH:M<br>M | DDMMMYYYY:HH:MM | DDMMMYYYY | XXX | No | Other | XXXXXX |
| XXXXX | XX/A4 | DDMMMYYYY | DDMMMYYYY:HH:M<br>M | DDMMMYYYY:HH:MM | DDMMMYYYY | | | | |

---

<sup>[1]</sup> Age in years; Race: A1 = African American/African Heritage, A2 = American Indian Or Alaskan Native, A3 = Asian-Central/South Asian Heritage, A4 = Asian-East Asian Heritage, A5 = Asian-Japanese Heritage, A6 = Asian-South East Asian Heritage, N = Native Hawaiian Or Other Pacific Islander, W1 = White-Arabic/North African Heritage, W2 = White - White/Caucasian/European Heritage, MT = Multiple.

<sup>[2]</sup> Duration in the study = (completion/withdrawal date and time - study product start date/time) + 1.

<sup>[3]</sup> Further details of reasons for withdrawal.


Protocol 207192 Program Run Date: DDMMYYYY

Listing 16.2.1.1.2 Subject Disposition All Non-Randomized Subjects

| Subject Number Age/Race [1] So | creening Date | Reason for Screen Failure | Further Details [2] |
|---|---|---|---|
| XXXXXX XX/A1 D | DDMMMYYYY | xxxxx | XXXXXX |

[1] Age in years; Race: A1 = African American/African Heritage, A2 = American Indian Or Alaskan Native, A3 = Asian-Central/South Asian Heritage, A4 = Asian-East Asian Heritage, A5 = Asian-Japanese Heritage, A6 = Asian-South East Asian Heritage, N = Native Hawaiian Or Other Pacific Islander, W1 = White-Arabic/North African Heritage, W2 = White - White/Caucasian/European Heritage, MT = Multiple.

[2] Further details of reasons for screen failure.

Program: xxxxxx.sas

Page x of y Source: Filename


Protocol 207192 Program Run Date: DDMMYYYY

Listing 16.2.2.1 Major Protocol Deviations All Randomized Subjects

Study Population: All Randomized Subjects(N=xx)

Product Group: XXXXXX

| Subject | Age/Race [1] | Visit(s)Excluded from PP Population | Deviation Reason |
|---|---|---|---|
| 10001 | 25/I | All From Visit 3 | Did not meet Inclusion criteria Did not meet Inclusion criteria Inclusion criteria |
| | | Visit 4 only | Treatment non-compliance |
| | | XX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | xx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |

<sup>[1]</sup> Age in years; Race: A1 = African American/African Heritage, A2 = American Indian Or Alaskan Native, A3 = Asian-Central/South Asian Heritage, A4 = Asian-East Asian Heritage, A5 = Asian-Japanese Heritage, A6 = Asian-South East Asian Heritage, N = Native Hawaiian Or Other Pacific Islander, W1 = White-Arabic/North African Heritage, W2 = White - White/Caucasian/European Heritage, MT = Multiple

Page x of y

Program: XXXXXXXXX.sas

Source: Filename

**Programming Note:** This listing is based on details in the population definition document.


Protocol 207192 Program Run Date: DDMMYYYY

Listing 16.2.2.2 Minor Protocol Deviations All Randomized Subjects

Study Population: All Randomized Subjects(N=xx)

Product Group: Test Product

| Subject Number | Age/Race [1] | Deviation Sequence | Start Date/Time of<br>Deviation | End Date/Time of<br>Deviation | Deviation Description |
|---|---|---|---|---|---|
| XXXXXX | XX/A1 | 1 | DDMMMYYYY:HH:MM | DDMMMYYYY:HH:MM | XXXXXX |

---

<sup>[1]</sup> Age in years; Race: A1 = African American/African Heritage, A2 = American Indian Or Alaskan Native,A3 = Asian-Central/South Asian Heritage, A4 = Asian-East Asian Heritage, A5 = Asian-Japanese Heritage, A6 = Asian-South East Asian Heritage, N = Native Hawaiian Or Other Pacific Islander, W1 = White-Arabic/North African Heritage, W2 = White - White/Caucasian/European Heritage, MT = Multiple


Protocol 207192 Program Run Date: DDMMYYYY

Listing 16.2.3.1
Exclusion from Analysis Populations
All Randomized Subjects

Study Population: All Randomized Subjects (N=xx) Product Group: Test Product

| Subject Number | Age/Race[1] | Safety Population | ITT Population | PP population |
|---|---|---|---|---|
| XXXXXX | XX/A1 | YES | YES | YES |

---

**Programming Note:** This listing is based on population definition document.


Protocol 207192 Program Run Date: DDMMYYYY

# Listing 16.2.4.1 Demographic and Baseline Characteristics All Randomized Subjects

#### Study Population: All Randomized Subjects(N=xx)

Product Group: Test Product

| Subject<br>Number | Age (years) | Sex | Race | Height (cm) | Weight (kg) | Body Mass Index<br>(kg/m²) | Stratification |
|---|---|---|---|---|---|---|---|
| XXXXXX | XX | Female | African American/African Heritage | xxx.x | XXX.X | XX.X | ≥ 25 - < 35 YEARS |
| XXXXXX | XX | Female | African American/African Heritage | xxx.x | XXX.X | XX.X | ≥ 35 - ≤ 45 YEARS |

Page x of y

Program: xxxxxx.sas Source: Filename


Protocol 207192 Program Run Date: DDMMYYYY

Listing 16.2.4.2 Medical History All Randomized Subjects

Study Population: All Randomized Subjects(N=xx)

Product Group: Test Product

| Subject Number | Age/Race[1] | Any Medical History | Medical Condition | Start Date | End Date or Ongoing |
|---|---|---|---|---|---|
| XXXXXX | XX/A1 | Yes | xxxxxx | DDMMMYYYY | DDMMMYYYY |
| xxxxxx | XX/A6 | Yes | XXXXXX | DDMMMYYYY | Ongoing |

[1] Age in years; Race: A1 = African American/African Heritage, A2 = American Indian Or Alaskan Native, A3 = Asian-Central/South Asian Heritage, A4 = Asian-East Asian Heritage, A5 = Asian-Japanese Heritage, A6 = Asian-South East Asian Heritage, N = Native Hawaiian Or Other Pacific Islander, W1 = White-Arabic/North African Heritage, W2 = White - White/Caucasian/European Heritage, MT = multiple

Program: xxxxxxx.sas Source: Filename


Protocol 207192 Program Run Date: DDMMYYYY

# Listing 16.2.5.1 Study Product Administration and Compliance All Randomized Subjects

Study Population: All Randomized Subjects (N=xx)

| D | ro | di i | ct | Gro | un. | Test | Prod | luct |
|---|----|------|----|-----|-----|------|------|------|

| Subject<br>Number | Age/Rac<br>e[1] | Visit | Date<br>Study<br>Product<br>Dispensed | Date/Time of<br>Product<br>Administered | Exposure<br>(in days)[2] | Number of<br>Sachets<br>Dispensed | Number of<br>Empty Sachets<br>Returned [3] | Number of<br>Uncomsumed<br>Sachets<br>Returned | Actual Number<br>of Sachets<br>Consumed [4] | Expected number of Sachets consumed[5] | Compliance<br>(%)[6] | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxx | XX/A1 | Baseline | DDMMM<br>YYYY | DDMMMYYYY:HH<br>:MM | | xxx | | | | | | |
| | | Visit 3 | DDMMM<br>YYYY | DDMMMYYYY:HH<br>:MM | х | xxx | xx | xx | x | x | 97 | |
| | | Visit 4 | DDMMM<br>YYYY | DDMMMYYYY:HH<br>:MM | x | xxx | xx | xx | x | x | 97 | |
| | | Visit 5 | DDMMM<br>YYYY | DDMMMYYYY:HH<br>:MM | x | xxx | xx | xx | x | x | 98 | |
| | _ | Visit 6 | DDMMM<br>YYYY | DDMMMYYYY:HH<br>:MM | x | xxx | xx | xx | x | x | 98 | |
| | = | Overall | | | | xxx | xx | xx | х | X | 98 | |

<sup>[1]</sup> Age in years; Race: A1 = African American/African Heritage, A2 = American Indian Or Alaskan Native, A3 = Asian-Central/South Asian Heritage, A4 = Asian-East Asian Heritage, A5 = Asian-Japanese Heritage, A6 = Asian-South East Asian Heritage, N = Native Hawaiian Or Other Pacific Islander, W1 = White-Arabic/North African Heritage, W2 = White - White/Caucasian/European Heritage, MT = multiple.

Page x of y

<sup>[2]</sup> Exposure = (Date/Time of Last Product Administered - Date/Time of First Product Administered)+1.

<sup>[3]</sup> As reported in eCRF.[4] actual number of sachets consumed = (number of sachets dispensed – number of sachets unconsumed returned)

<sup>[5]</sup> Expected number of sachets consumed = 2 sachets\*Number of days between the visits.

<sup>[6]</sup> By Visit Compliance = (Actual number of sachets consumed / expected number of sachets consumed) \* 100; Overall compliance = (actual total number of sachets consumed / expected total number of sachets consumed)

<sup>\*</sup> Subjects with compliance > 120% or less than 80%.

| Fortified | HFD |
|-----------|-----|
| 207192 | |


Program: xxxxxx.sas Source: Filename

**Programming Note:** Overall compliance will not be calculated for the subjects who discontinued before completing visit 6 Highlight compliance values with '\*' if the compliance is more than 120% or less than 80%.


Protocol 207192 Program Run Date: DDMMYYYY

Listing 16.2.5.2 Prior Medications All Randomized Subjects

Study Population: All Randomized Subjects(N=xx)

Product Group: Test Product

Program: xxxxxx.sas

| Subject<br>Number | Age/Race[1] | Sequence<br>Number | Drug Name<br>[GSK Drug Synonym] | Reason for<br>Medication | Route of Admin. | Dose per Admin.<br>(unit) | Frequency | Start Date<br>(Study Day [2]) | End Date/ Ongoing |
|---|---|---|---|---|---|---|---|---|---|
| | | Nullibei | | | | , , | | | |
| XXXXXX | XX/A6 | 1 | [XXXXXX] | XXXXXX | XXXXXX | XXXXXX (xx) | XXXXXX | DDMMMYYYY<br>(XX) | Ongoing |
| XXXXXX | XX/A6 | 1 | XXXXXX<br>[XXXXXX] | XXXXXX | XXXXXX | XXXXXX (xx) | xxxxx | DDMMMYYYY<br>(XX) | DDMMMYYYY |

Page x of y
Source: Filename

**Programming Note:** Similar listing will be generated for Concomitant Medications and Non-Drug Therapies.

<sup>[1]</sup> Age in years; Race: A1 = African American/African Heritage, A2 = American Indian Or Alaskan Native, A3 = Asian-Central/South Asian Heritage, A4 = Asian-East Asian Heritage, A5 = Asian-Japanese Heritage, A6 = Asian-South East Asian Heritage, N = Native Hawaiian Or Other Pacific Islander, W1 = White-Arabic/North African Heritage, W2 = White - White/Caucasian/European Heritage, MT=Multiple.
[2] Study day relative to the date of first dose of treatment.


Protocol 207192 Program Run Date: DDMMYYYY

## Listing 16.2.6.1 Serum Type I Collagen CrossLinking C-Telopeptide All Randomized Subjects

Study Population: All Randomized Subjects(N=xx)

Product Group: Test Product
Normal Range (xx x - xx x)

| Subject Number | Age/Race<br>[1] | Visit | Date of Visit | Was Assessment<br>Performed? | Date of Sample<br>Collection/Time of Sample<br>Collection | Sample<br>Assessment Date | Result (unit) | Change<br>from<br>Baseline | Comment |
|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | XX/N | Screening<br>Baseline | DDMMMYYYY<br>DDMMMYYYY | Yes | DDMMMYYYY/hh:mm | DDMMMYYYY | xx.x<br>xx.x | | xxx<br>xxxx |
| | | Visit 5<br>Visit 6 | DDMMMYYYY<br>DDMMMYYYY | Yes | DDMMMYYYY/hh:mm | DDMMMYYYY | xx.x | xx.x<br>xx.x | xxxxx |

---

[1] Age in years; Race: A1 = African American/African Heritage, A2 = American Indian Or Alaskan Native, A3 = Asian-Central/South Asian Heritage, A4 = Asian-East Asian Heritage, A5 = Asian-Japanese Heritage, A6 = Asian-South East Asian Heritage, N = Native Hawaiian Or Other Pacific Islander, W1 = White-Arabic/North African Heritage, W2 = White - White/Caucasian/European Heritage, MT=Multiple.

Program: xxxxxxx.sas Source: Filename

#### **Programming Note:**

- Repeat the same layout for listing 16.2.6.2-16.2.6.19 and 16.2.6.22
- For the following laboratory tests normal ranges will not be displayed Serum Cross-Linked C-Telopeptide of Type 1 Collagen, Ratio of Carboxylated to Under-Carboxylated Osteocalcin, Urinary C-Telopeptide of Type 1 Collagen, Serum Vitamin D (using 25-OH D3), Urinary Calcium/Creatinine Ratio and Serum Folate


Protocol 207192 Program Run Date: DDMMYYYY

Listing 16.2.6.20
Listing of Normal Range for Blood and Urine Parameters

| Parameter (Unit) | Biological Matrix | Gender | Age Range (in years) | Normal | Range |
|---|---|---|---|---|---|
| | | | | Lower Limit | Upper Limit |
| Serum Type I Collagen Cross-<br>linked C-telopeptide (unit) | Blood | Male | XX-XX | | |
| | | Female | xx-xx | | |
| | | | | | Page x of y |
| Program: xxxxxx.sas | | | Source: Filename | | |


Protocol 207192 Program Run Date: DDMMYYYY

#### Listing 16.2.6.21 Seven Day Dietary Intake Assessment All Randomized Subjects

Study Population: All Randomized Subjects (N=xx)

| Product Group: | lest | Proc | luct |
|----------------|------|------|------|
|----------------|------|------|------|

| Subject | Age/Race[1 | Visit | Date of Visit | Total Energy (Kcal) | | | | | | Average Sele | enium intake (mcg) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Number | J | | | Observed value | Change<br>from | Observed value | Change<br>from | Observed value | Change<br>from | Observed value | Change from<br>Baseline |
| | | | | | Baseline | | Baseline | | Baseline | | |
| | | Screening | DDMMMYYYY | | | | | | | | |

[1] Age in years; Race: A1 = African American/African Heritage, A2 = American Indian Or Alaskan Native, A3 = Asian-Central/South Asian Heritage, A4 = Asian-East Asian Heritage, A5 = Asian-Japanese Heritage, A6 = Asian-South East Asian Heritage, N = Native Hawaiian Or Other Pacific Islander, W1 = White-Arabic/North African Heritage, W2 = White - White/Caucasian/European Heritage, MT=Multiple.

Source: Filename

Page x of y

Program: xxxxxx.sas

**Programming Note:** This listing will include all parameters for dietary intake assessment [Total Energy intake (Kcal), Total Carbohydrate intake (gm), Total Fat intake (gm), Average Calcium intake (mg), Average protein intake (g), Average Vitamin D intake (mcg), Average Vitamin B6 intake (mg), Average Vitamin B12 intake (mg), Average Phosphorous intake (mg), Average Folic Acid intake (mcg), Average Zinc intake (mg), and Average Selenium intake (mcg)].


Protocol 207192 Program Run Date: DDMMYYYY

Listing 16.2.7.1.1 All Adverse Events All Randomized Subjects

Study Population: All Randomized Subjects(N=xx)

Product Group: Test Product

| acc c. capc. | 5064460 | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Age/Race[1] | Adverse Event<br>(Preferred Term)<br>[System Organ Class] | Start Date/Time/ Study Day[2] | End Date/<br>Time | Frequency/<br>Intensity | Related to<br>Study<br>Product? | Action Taken<br>with Study<br>Product | Outcome | Serious? | Subject<br>Withdrawn |
| xxxxxx | XX/N | HEADACHE<br>(NERVOUS SYSTEM<br>DISORDER)<br>[xxxxxxxx] | 31MAR2017/<br>HH:MM:SS/<br>3 | DDMMMYYYY/<br>HH:MM:SS | SINGLE<br>EPISODE/<br>MILD | No | NOT<br>APPLICABLE | RECOVERED/<br>RESOLVED | NO | NO |

[1] Age in years; Race: A1 = African American/African Heritage, A2 = American Indian Or Alaskan Native, A3 = Asian-Central/South Asian Heritage, A4 = Asian-East Asian Heritage, A5 = Asian-Japanese Heritage, A6 = Asian-South East Asian Heritage, N = Native Hawaiian Or Other Pacific Islander, W1 = White-Arabic/North African Heritage, W2 = White - White/Caucasian/European Heritage.
[2] Study day is the day relative to start of treatment.

Page x of y

Program: xxxxxx.sas Source: Filename

Programming Note for Listing 16.2.7.1.2:

- Repeat the same layout for listing 16.2.7.1.2
- Population should be used 'Non randomized Subjects'
- The fourth column should be only 'Start Date/Time (take out Study Day)'


# Fortified HFD 207192 Final Statistical Reporting and Analysis Plan Addendum Version 2.0 23-July-2018 • Delete the footnote related to study day and adjust the numbers accordingly.


Protocol 207192 Program Run Date: DDMMYYYY

Listing 16.2.9.1 Vital Signs All Randomized Subjects

Study Population: All Randomized Subjects(N=xx)

Product Group: Test Product

| Subject | Age/Race[1 | Visit | Date of Visit | Date of | Systolic Blood Pressure (mmHg) | | Diastolic Blood<br>Pressure (mmHg) | | Heart<br>Rate (beats/min) | | Oral Temperature (F) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Number | 1 | | | Assessment | | | | | | | | |
| | | | | | Observed | Change | Observed | Change | Observed | Change | Observed | Change from |
| | | | | | value | from | value | from | value | from | value | Baseline |
| | | | | | | Baseline | | Baseline | | Baseline | | |
| | | Screening | DDMMMYYY | DDMMMYYYY | | | | | | | | |
| | | _ | V | | | | | | | | | |

<sup>[1]</sup> Age in years; Race: A1 = African American/African Heritage, A2 = American Indian Or Alaskan Native, A3 = Asian-Central/South Asian Heritage, A4 = Asian-East Asian Heritage, A5 = Asian-Japanese Heritage, A6 = Asian-South East Asian Heritage, N = Native Hawaiian Or Other Pacific Islander, W1 = White-Arabic/North African Heritage, W2 = White - White/Caucasian/European Heritage, MT=Multiple.

Page x of y
Program: xxxxxxx.sas Source: Filename


Protocol 207192 Program Run Date: DDMMYYYY

Listing 16.2.9.2 Physical Examination All Randomized Subjects

Study Population: All Randomized Subjects(N=xx)

Product Group: Test Product

| Subject Number | Age/Race[1] | Visit | Date of Visit | Body System | Finding | Description of Abnormality, CS or Not<br>Examined |
|---|---|---|---|---|---|---|
| xxxxxx | xx/n | Screening | DDMMMYYYY | CNS<br>Eyes<br>ENT<br>Respiratory | Normal<br>Normal<br>Abnormal, CS<br>Normal | xxxxxx |

<sup>[1]</sup> Age in years; Race: A1 = African American/African Heritage, A2 = American Indian Or Alaskan Native, A3 = Asian-Central/South Asian Heritage, A4 = Asian-East Asian Heritage, A5 = Asian-Japanese Heritage, A6 = Asian-South East Asian Heritage, N = Native Hawaiian Or Other Pacific Islander, W1 = White-Arabic/North African Heritage, W2 = White - White/Caucasian/European Heritage, MT=Multiple.

Programming Note for Listing 16.2.9.2: If subjects has abnormality description and CS description, please concatenate both separating with ','.


Protocol 207192 Program Run Date: DDMMYYYY

Listing 16.2.9.3 Hemoglobin Assessment All Randomized Subjects

Study Population: All Randomized Subjects(N=xx)

Product Group: Test Product

| Subject<br>Number | Age/Race<br>[1] | Visit | Date of Visit | Was Hb<br>Assessment<br>Performed?[2<br>] | Hb Assessment Results (g/dL) | |
|---|---|---|---|---|---|---|
| | | | | | Observed value | Change from<br>Baseline |
| xxxxx | XX/N | Screening<br>Baseline | DDMMMYYYY<br>DDMMMYYYY | Yes | XX.X<br>XX.X | xx.x<br>xx.x |
| | | Visit 5<br>Visit 6 | DDMMMYYYY<br>DDMMMYYYY | Yes | | xx.x<br>xx.x |

<sup>[1]</sup> Age in years; Race: A1 = African American/African Heritage, A2 = American Indian Or Alaskan Native, A3 = Asian-Central/South Asian Heritage, A4 = Asian-East Asian Heritage, A5 = Asian-Japanese Heritage, A6 = Asian-South East Asian Heritage, N = Native Hawaiian Or Other Pacific Islander, W1 = White-Arabic/North African Heritage, W2 = White - White/Caucasian/European Heritage, MT=Multiple. [2] Yes = Assessment performed; No = Assessment not done.

Program: xxxxxxx.sas Source: Filename


Protocol 207192 Program Run Date: DDMMYYYY

Figure 14.2.2.1 Serum Cross Linked C-Telopeptide of Type 1 Collagen Least Square Mean(  $\pm$ -SE) by Time and Treatment ITT Population



Program: xxxxxx.sas Source: Filename

Programming Note: All other figures will follow the same format. Use one solid line and one dotted line for each treatment. LSMEANS and SE will be obtained from Table 14.2.2.2. Baseline will obtained from the raw values. X-axis will be labeled for baseline, 3 Month and 6 Month.